Amgen Protocol #: 20139075

# TITLE: Neoadjuvant Intralesional Injection of Talimogene Laherparepvec with Concurrent Preoperative Radiation in Patients with Locally Advanced Soft Tissue Sarcomas

**Coordinating Center:** Holden Comprehensive Cancer Center – University of Iowa.

\*Principal Investigator: Mohammed Milhem, MD

Clinical Professor

Department of Internal Medicine, Division

of Medical Oncology

C-32 GH 319-356-2324

mohammed-milhem@uiowa.edu

# **Co-Investigators:**

Carryn Anderson, MD
Clinical Assistant Professor
Department of Radiation Oncology
University of Iowa Hospitals and Clinics
01612D PFP
(319) 353-8836
carryn-anderson@uiowa.edu

Varun Monga, M.D.
Clinical Assistant Professor
Division of Hematology, Oncology, &
Blood and Marrow Transplantation
Department of Internal Medicine
University of Iowa Hospitals and Clinics
C-32 GH
(319) 384-9497
varun-monga@uiowa.edu

Benjamin J. Miller, MD Assistant Professor Department of Orthopedic Surgery University of Iowa Hospitals and Clinics 01008 JPP (319) 356-2488 benjamin-j-miller@uiowa.edu

Bryan Allen, MD, PhD Associate Professor Department of Radiation Oncology 200 Hawkins Drive, Iowa City, IA 52242 (319) 353-8836 bryan-allen@uiowa.edu Munir Tanas, MD Assistant Professor Department of Surgical Pathology University of Iowa Hospitals and Clinics 1026 ML (319) 335-6637 munir-tanas@uiowa.edu

#### **Correlative Study Team**

Steven Varga, PhD Professor of Microbiology and Immunology Professor of Pathology 205 Gilmore Hall, Iowa City, Iowa 52242

Office: 319-353-2361

Weizhou Zhang, PhD University of Florida Department of Pathology and Immunology 1333 Center Drive, BG-022b Gainesville, FL 32610-0275

#### Biostatistician

Sarah Bell, MS Holden Comprehensive Cancer Center 145 N Riverside Dr, N319 CPHB | Iowa City, IA 52242 Email: <a href="mailto:sarah-mott@uiowa.edu">sarah-mott@uiowa.edu</a> | Cell: 319-217-0376

**Study Agent:** Talimogene Laherparepvec

Other Agent(s): Standard external beam radiation

| Investigational Agent | IND# | IND Sponsor |
|--------------------------|-------|-----------------|
| Talimogene Laherparepvec | 16359 | Mohammed Milhem |

Protocol #: 20139075 Protocol Version Date: 4/8/2014

Amendment 1: 1/13/2014 Amendment 2: 4/8/2014 Amendment 3: 7/21/2014 Amendment 4: 7/25/2014 Amendment 5: 12/15/2014 Amendment 6: 3/30/2015 Amendment 7: 9/13/2015 Amendment 8: 10/26/2015 Amendment 9: 3/17/2016 Amendment 10: 11/15/2016 Amendment 11: 12/22/2017 Amendment 12: 6/24/2020 Amendment 12.1: 10/9/2020 Amendment 13: 3/21/2021 Amendment 14: 4/21/2021 Amendment 15: 10/17/2022

Amendment 15.1: 3/13/2023

#### **SCHEMA**

# **Study Timeline Schema:**



# Phase 1b schema:



Table 1. Phase 1b Dose De-escalation Schedule

| Number of Patients with DLT at a | Decision Rule |
|---|---|
| Given Talimogene Laherparepvec | |
| Dose | |
| $\geq 2$ | Dose level will be declared toxic. |
| | If this is the lowest dose level, stop the study due to |
| | excessive toxicity; otherwise enter three additional |
| | patients at the next lowest dose level. |
| $\leq 1$ out of 3 | Enter <i>three</i> more patients at this dose level. |
| $\leq 1$ out of 6 | This is the recommended Phase II dose. |

# **Talimogene Laherparepvec Dose Levels:**

Dose 0 = talimogene laherparepvec up to 8.0 mL of 10<sup>8</sup> PFU/mL dosed weekly Dose -1 = talimogene laherparepvec up to 8.0 mL of 10<sup>8</sup> PFU/mL dosed every 2 weeks.

• Initial dose for all = talimogene laherparepvec up to 4.0 mL of 10<sup>6</sup> PFU/mL

# Phase 2 Schema:



# **TABLE OF CONTENTS**

| SCH | HEMA | 3 |
|---|---|---|
| 1. | BACKGROUND | 7<br>7<br>10 |
| 2. | REGISTRATION PROCEDURES | |
| 3. | OBJECTIVES | 12 |
| 4. | PATIENT SELECTION | 13 |
| 5. | TREATMENT PLAN AND STUDY SCHEMA 5.1 Study Design 5.2 Study Agent Administration: Talimogene Laherparepvec 5.3 General Concomitant Medication and Supportive Care Guidelines 5.4 Duration of Therapy 5.5 Duration of Follow Up 5.6 Criteria for Removal from Study | 16<br>23<br>23<br>23 |
| 6. | DOSING DELAYS/DOSE MODIFICATIONS. 6.1 Dose Delays 6.2 Dose Limiting Toxicities 6.3 Dose Reductions | 25 |
| 7. | ADVERSE EVENTS: LIST AND REPORTING REQUIREMENTS 7.1 Adverse Event Definitions 7.2 Adverse Event Characteristics 7.3 Comprehensive Adverse Events and Potential Risks List (CAEPR) 7.4 Important Potential Risks 7.5 PREGNANCY AND BREASTFEEDING 7.6 Other Relevant Information 7.7 Expedited Adverse Event Reporting | 27<br>28<br>30<br>33 |
| 8. | PHARMACEUTICAL INFORMATION | |
| 9. | CORRELATIVE, AND SPECIAL STUDIES | 40 |
| 10. | STUDY CALENDAR | |

| NCI I | Protocol | #: | |
|-------|----------|-----------------------------------------|----|
| Versi | on Date: | March, 13, 2023 | |
| | 10.2 | Screening Procedures | 43 |
| | 10.3 | Long-term Follow up | 43 |
| 11. | MEAS | SUREMENT OF EFFECT | 44 |
| | 11.1 | Pathologic Response | 44 |
| | 11.2 | Time to Disease progression (TTP) | 44 |
| | 11.3 | Other Response Parameters | |
| 12. | STAT | ISTICAL CONSIDERATIONS | 45 |
| | 12.1 | Study Design/Endpoints | 45 |
| REFI | ERENCE | S | 46 |
| APPI | ENDIX A | PERFORMANCE STATUS CRITERIA | 49 |
| APPI | ENDIX I | RECIST GUIDELINES | 50 |
| APPI | ENDIX ( | C: CTCAE v.4.0 | 51 |
| APPI | ENDIX I | D: CONTRAINDICATIONS AND ADVERSE EVENTS | 52 |
| • | Routi | ne Adverse Event Reporting | 56 |
| • | Serio | us Adverse Event Reporting | 57 |

#### 1. BACKGROUND

# 1.1 Disease Background

Adult soft tissue sarcomas (STS) constitute a wide heterogeneous group of very rare tumors, both in terms of histology and biological and clinical behavior. In contrast to major advances in the biological understanding of these heterogeneous subtypes, forward progress in the systemic treatment of sarcoma has been painstakingly slow. The prognosis of patients with metastatic or recurrent disease is poor and most of them will die from tumor progression. Taking into account differences in histology subtype, anatomic location of disease and age at disease onset, the overall median survival for patients with metastatic STS is approximately one year and only about 10% of these patients are alive at five years.<sup>1</sup>

Control of localized disease is, therefore, of prime importance as evidenced by the National Comprehensive Cancer Network's (NCCN) current treatment guidelines.<sup>2</sup> Pisters et al demonstrated that histologic grade, depth of location, and positive surgical margins are key determinants of STS recurrence.<sup>3</sup> However, patients typically present late with local tumor extensions into critical adjacent structures, making complete surgical resection with uninvolved margins difficult. Preoperative radiotherapy has been shown to significantly improve local disease control, functional outcomes and survival in patients with locally advanced STS.<sup>4-6</sup>

#### 1.2 Talimogene Laherparepvec

Talimogene laherparepvec (HSV-1 [strain JS1]/ICP34.5-/ICP47-/hGM-CSF) is an oncolytic immunotherapy, formerly known as OncoVEX<sup>GM-CSF</sup>, an immune-enhanced, oncolytic herpes simplex virus type 1 (HSV-1). Talimogene laherparepvec is a replication-competent HSV-1 designed for intratumoral injection. Talimogene laherparepvec was constructed using a new isolate of HSV-1 (strain JS1; ECACC Accession Number 01010209) and has been sequenced. The neurovirulence factor ICP34.5 and the ICP47-encoding genes are functionally deleted in the virus. The ICP34.5 functional deletion allows the virus to replicate selectively in tumors. The role of ICP47 is to block antigen presentation to major histocompatibility complex (MHC) class I and II molecules by blocking the transporter associated with antigen processing 1 and 2 (TAP1, TAP2). This deletion also allows the increased expression of the US11 gene. This promotes virus growth in cancer cells without decreasing tumor selectivity. The virus contains the coding sequence for human GM-CSF, a pleotropic cytokine involved in the stimulation of cellular immune responses.

Development of talimogene laherparepvec was conducted in conjunction with the International Conference on Harmonization (ICH) guidance on oncolytic viruses. The therapeutic strategy for talimogene laherparepvec is to effect tumor cell death by lytic virus replication following direct intratumoral injection, combined with induction of an anti-tumor immune response enhanced by the local expression of GM-CSF. This combination of direct lysis of the injected tumor plus enhancement of the patient's own immune response is intended to result in both local and distant tumor destruction, and to prevent future progression of disease.

Version Date: March, 13, 2023

The preparation and testing of the cell banks, viral seed stock, and talimogene laherparepvec clinical material were conducted in accordance with current Good Manufacturing Practices (cGMP), relevant ICH guidelines, European Directives, and the US Pharmacopeia and Title 21 Code of US Federal Regulations. In particular, the European Pharmacopoeia (Ph Eur) monograph on viral vaccine testing, ICH considerations on Oncolytic Viruses, and Food and Drug Administration (FDA) Points to Consider – Characterization of Cell Lines Used to Produce Biologicals (1993) have been followed for the safety testing of talimogene laherparepvec.

Talimogene laherparepvec has been studied in several clinical trials in multiple tumor types. A summary of talimogene laherparepvec's pertinent efficacy results and safety data follow. After intra-tumoral injection, talimogene laherparepvec is generally cleared from subjects' blood and urine within 48 hours. Rarely, extremely low levels of virus have been detected on the surface of injected tumors for up to 2 weeks following a single dose. In most cases, this was observed in seronegative subjects in the phase 1 study, in which a higher first dose of talimogene laherparepvec was administered than has been used in subsequent studies. Subsequent studies have therefore used a lower initial dose (see below). No evidence of herpes infection attributable to talimogene laherparepvec has been documented in study subjects. While a number of individuals (subjects or medical personnel) have had reactivations of wild type HSV-1, which is not unexpected in the population as a whole, it was determined by culture of the virus and polymerase chain reaction (PCR) analysis not to be caused by talimogene laherparepvec.

Please refer to the talimogene laherparepvec Investigator Brochure (IB) for descriptions of all available data.

# 1.2.1 Talimogene Laherparepvec Clinical Experience

Nine clinical studies have been or are being conducted in several advanced tumor types including advanced solid tumors, melanoma, squamous cell cancer of the head and neck, and pancreatic cancer.<sup>28</sup>

These studies include a phase 1 study to evaluate the safety, bio-distribution, and biological activity of differing dose levels of talimogene laherparepvec in patients with advanced solid tumors. <sup>27</sup> In this open-label, ascending-dose study, single doses of talimogene laherparepvec either 10<sup>6</sup>, 10<sup>7</sup>, or 10<sup>8</sup> plaque forming units/mL (PFU/mL) (up to 4 mL), were injected directly into a single metastatic skin or subcutaneous tumor of breast cancer, head and neck cancer, gastrointestinal cancer, or melanoma. This study, as reported by Hu et al, identified that subjects who are seronegative for HSV-1 more commonly developed febrile flu-like symptoms and erythematous skin rashes at higher initial doses of talimogene laherparepvec (10<sup>7</sup> and 10<sup>8</sup> PFU/mL) compared to a decreased initial dose of 10<sup>6</sup> PFU/mL. <sup>27</sup>

In a phase I/II upward-titration study to assess the safety and biological activity of three dose levels of talimogene laherparepvec (all initial doses were 10<sup>6</sup> PFU/mL, followed by subsequent doses of 10<sup>6</sup>, 10<sup>7</sup> or 10<sup>8</sup> PFU/mL) a greater mean decrease in tumor size was observed in patients receiving subsequent doses of 10<sup>7</sup> PFU/mL or higher compared to those administered only 10<sup>6</sup> PFU/mL for all doses. The study also reported that none of the injected tumors in the lowest dose cohort (10<sup>6</sup> PFU/mL) had resolved by the end of the treatment period, whereas 36.5%


(12/32) of measurable tumors resolved (i.e., were no longer detectable) at the higher dose levels, suggesting that talimogene laherparepvec has a dose-related effect on tumor necrosis. <sup>26</sup> Necrosis of injected tumors, confirmed on histopathology, was observed in both seropositive and seronegative subjects. These data supported the conclusion that an initial dose of 10<sup>6</sup> PFU/mL, followed by doses of 10<sup>8</sup> PFU/mL, was appropriate for use in further trials. This dose regimen has been used in several ongoing phase III of trials including in subjects with advanced stage melanoma. <sup>28</sup>

Clinical data currently available indicate that talimogene laherparepvec has the potential to provide overall clinical benefit to patients with advanced melanoma (Talimogene Laherparepvec Investigator's Brochure, 2012). In particular, a high rate of complete response (CR) was achieved (20% in the phase 2 study with talimogene laherparepvec in stage IIIc to IV melanoma). Response was still ongoing for all but 1 subject at the time of the last tumor evaluation, with a median duration of longest response of 223 days (Talimogene Laherparepvec Investigator's Brochure, 2012). In addition, responses were observed in both injected and uninjected sites, including visceral sites.

In another study, patients with stage III/IVA/IVB squamous cell cancer of the head and neck (SCCHN) were treated with intra-tumoral injections of talimogene laherparepvec in combination with chemoradiotherapy in a phase I/II study. Subjects received chemoradiotherapy (70 Gy/35 fractions with concomitant cisplatin 100 mg/m2 on days 1, 22, and 43) and dose-escalating (10<sup>6</sup>, 10<sup>6</sup>, 10<sup>6</sup>, 10<sup>6</sup> pfu/mL for cohort 1; 10<sup>6</sup>, 10<sup>7</sup>, 10<sup>7</sup>, 10<sup>7</sup> for cohort 2; 10<sup>6</sup>, 10<sup>8</sup>, 10<sup>8</sup>, 10<sup>8</sup> for cohort 3) by intratumoral injection on days 1, 22, 43, and 64. Patients underwent neck dissection 6 to 10 weeks later.

The results from this study are reported in Harrington et al and indicate that seventeen patients were treated without delays to chemoradiotherapy or dose-limiting toxicity. Fourteen patients (82.3%) showed tumor response by Response Evaluation Criteria in Solid Tumors, and pathologic complete remission was confirmed in 93% of patients at neck dissection. HSV was detected in injected and adjacent uninjected tumors at levels higher than the input dose, indicating viral replication. All patients were seropositive at the end of treatment. No patient developed locoregional recurrence, and disease-specific survival was 82.4% at a median follow-up of 29 months (range, 19-40 months).<sup>26</sup>

Recently a Phase 1b/2 trial using Talimogene Laherparepvec in locally advanced soft tissue sarcomas was completed at University of Iowa. A total of 30 subjects were enrolled. No dose limiting toxicities were observed with the 4 mL dose containing 10<sup>8</sup> PFU/mL. 24% patients achieved 95% pathological necrosis (*verbal communication, manuscript submitted*). The proposed primary endpoint of 30% patients with 95% path necrosis was not reached. One of the possibilities for failure to reach this endpoint was the inadequate drug distribution relative to the size of these tumors. Hence a new trial with higher amount of injectable drug is being proposed.

#### 1.2.2 Talimogene Laherparepvec Safety Experience


An observational registry study is ongoing to investigate the long-term survival and safety of subjects previously treated with talimogene laherparepvec in any study. Preliminary safety data from the completed clinical studies for which adverse event data are available has shown that the most commonly ( $\geq 10\%$ ) occurring adverse events (without regard to causality and including talimogene laherparepvec given in combination with cisplatin and radiation) are nausea, vomiting, diarrhea, chills, pyrexia, fatigue, flu-like symptoms, injection site reactions, and myalgia. Other common ( $\geq 1\%$  and < 10%) reactions include arthralgia, pain in extremity, cellulitis, headaches, and dizziness. The adverse event profile, therefore, may include events related to talimogene laherparepvec, chemotherapy, radiation, tumor-related signs and symptoms, disease progression, and/or a combination of these. Data thus far supports talimogene laherparepvec to be a safe and well tolerated immunotherapy in human subjects.

#### Injection Site Reactions

Talimogene laherparepvec is administered by direct injection into cutaneous, subcutaneous, and nodal tumor masses. Injection site adverse events may occur, such as erythema, local skin discoloration, induration, warmth, and pain. Infrequently, injected cutaneous tumor masses may undergo necrosis, predisposing the subject to local and/or systemic infections. Similarly, injected pathologic lymph nodes may enlarge or become necrotic. Uncommonly, necrotic lymph nodes may be the site of persistent drainage that requires corrective measures. In clinical studies, adverse events of "injection site pain" and "injection site reaction" were very common, occurring in  $\geq 10\%$  of talimogene laherparepvec-treated subjects. Most events of injection site pain and injection site reaction in subjects receiving talimogene laherparepvec were mild to moderate in severity. Subjects seronegative at baseline for HSV-1, when given an initial dose of talimogene laherparepvec at a concentration of  $10^6$  PFU, do not appear to experience more exaggerated injection site reactions than those who are seropositive at baseline.

#### Cellulitis

Necrosis of cutaneous tumor masses and pathologic lymph nodes injected with talimogene laherparepvec may infrequently occur, predisposing to local/regional infection (ie, cellulitis). In clinical studies to date, cellulitis was common, occurring in  $\geq 1\%$  to < 10% of subjects treated with talimogene laherparepvec.

#### Flu-like Symptoms

Constitutional symptoms including chills, fatigue, headache, myalgia, and pyrexia may occur with talimogene laherparepvec. Collectively, this constellation of symptoms may be described as "flu-like symptoms." In clinical studies to date, adverse events with the MedDRA preferred terms "chills," "fatigue," "headache," "influenza like illness," "myalgia," and "pyrexia" were very common, occurring in  $\geq 10\%$  of subjects treated with talimogene laherparepvec. Most of these events were mild to moderate in severity. Subjects seronegative at baseline for HSV-1, when given an initial dose of talimogene laherparepvec at a concentration of  $10^6$  PFU, do not appear to experience more flu-like symptoms than those who are seropositive at baseline. These symptoms are self-limiting and resolve without sequelae.

#### 1.3 Radiation Therapy in Sarcoma

The benefits of combination therapy with radiation and surgery in significantly improving local

control in STS patients are well documented. Preoperative radiotherapy has been shown to significantly improve local disease control, functional outcomes and survival in patients with locally advanced STS. 4-6 Recent review of literature indicates that about 10% of patients will have  $\geq 95\%$  tumor necrosis, and about 25% will achieve  $\geq 80\%$  tumor necrosis following preoperative radiation therapy alone. 7-8 Further review indicates that only those patients who achieve  $\geq 95\%$  tumor necrosis with preoperative radiation have improved local and distant control as well as overall survival. Despite its reported benefits, radiotherapy is associated with a high rate of complications and significant functional morbidity. O'Sullivan et al compared preoperative versus postoperative external beam radiation (EBRT) for resectable extremity STS. Long term follow up revealed no statistical difference in local control and cause specific survival, however, preoperative radiotherapy was associated with a significantly higher rate of acute wound complications (35% vs. 17%, p = 0.01) and a lower rate of late Grade 2–4 fibrosis  $(32\% \text{ vs. } 48\%, p = 0.07).^{9-10}$  Multiple retrospective reviews have similarly found high rates of acute wound complications in sarcoma patients ranging from 25% to 44%. 11-14 These reported high rates of acute and late toxicities support the need for additional research to improve the safety profile of neoadjuvant radiotherapy.

In addition, there is need to improve efficacy of the radiation treatments to achieve higher rates of tumor necrosis, and, to ensure resection of the tumor with clear margins for successful organ preserving treatment of sarcoma.

#### 1.4 Rationale

Immunotherapy has long been discussed as a promising method for the treatment of patients with solid tumors but thus far its exact role in sarcoma remains to be defined. Analysis of sera from sarcoma patients indicate the presence of both humoral and cellular immune responses against cancer-testis antigens commonly associated with sarcoma tumors and sarcoma cell lines, indicating that immune modulation may play a central role in sarcoma-genesis. 15-17 Viruses have been used in the treatment of cancer since the early 20<sup>th</sup> century. <sup>16</sup> Herpes simples virus type 1 (HSV-1) is a highly lytic virus which infects a wide variety of human cell types and rapidly replicates itself, resulting in cell lysis and inflammation. This replication can be rendered tumor selective through deletion of the HSV-1 gene encoding ICP34.5. 19-20 Talimogene laherparenvec. is a replication-competent, immune-enhanced HSV-1 for intratumoral injection. It is made from a new HSV-1 strain in which the neurovirulence genes encoding ICP34.5 and ICP47 have been deleted. The deletion of ICP34.5 allows for selective replication of the virus in tumor cells. Deletion of ICP47 prevents the inhibition of antigen presentation usually caused by the expression of this protein, and also promotes tumor-selective viral replication. In addition, the ICP34.5-gene has been replaced with the coding sequence for human granulocyte macrophage colony stimulating factor (GM-CSF), to enhance the immune response to tumor antigens released from virus replication.<sup>21-22</sup>

The primary goal of this study is to improve on the 10% of patients who achieve  $\geq$  95% tumor necrosis historically seen with radiation therapy alone. Theoretically, replicating HSV-derived oncolytic agents are sufficient to cause impressive cell killing independent of any interactions with the immune system. Oncolytic HSV-1 elicits an immune response both to the HSV and to

tumor-specific antigens. The expressed GM-CSF further stimulates a cytotoxic T cell response against tumor antigens released through viral oncolysis. The T-cell stimulation index and the level of immune response may have important correlation with clinical vaccine efficacy, as seen in the phase III trial by Small et al. Additionally, there is growing evidence that radiation induces immunogenic tumor cell death and alters the tumor microenvironment to enhance recruitment of antitumor T cells and, thus, enhancing the overall immune response.

Finkelstein et al recently demonstrated enhanced antitumoral immune response following concurrent administration of dendritic cells and radiation compared to either therapy alone.<sup>23</sup> Similarly, synergistic effect between talimogene laherparepvec injection and radiotherapy has been reported in melanoma patients. <sup>24-26</sup> The efficacy and safety of talimogene laherparepvec is most mature in studies involving patients with malignant melanoma, pancreatic, and head and neck cancers. At least nine clinical trials and extended protocols have been or are being conducted with over 400 subjects treated with talimogene laherparepvec. <sup>24-28</sup> An observational registry study is ongoing to investigate the long-term survival and safety of subjects previously treated with talimogene laherparepvec in any study.<sup>27</sup> The most commonly ( $\geq 10\%$ ) reported adverse reactions are nausea, vomiting, diarrhea, chills, pyrexia, fatigue, flu-like symptoms, injection site reactions, and myalgia. Other common (> 1% and < 10%) reactions include arthralgia, pain in extremity, cellulitis, headaches, and dizziness. Concurrent therapy with talimogene laherparepvec, cisplatin, and EBRT in a recent phase II study was well tolerated and the adverse events were mostly mild (Grades 1 and 2). The most frequent toxicities and severity in this study were consistent with that seen with conventional chemoradiotherapy. <sup>26</sup> Data thus far supports talimogene laherparepvec to be a safe and well tolerated immunotherapy in human subjects.

#### 2. REGISTRATION PROCEDURES

All studies that undergo PRMC review and/or utilize HCCC Clinical Research Services (CRS) resources are required to register subjects in OnCore. Each subject registration includes the following:

- The subject's IRB approved (version date) consent form and the date of their consent.
- Date of eligibility and eligibility status (eligible, not eligible)
- On study date and subject's disease site (and histology if applicable)
- On treatment date (if applicable)

All subject registration information is expected to be entered into OnCore within **2 (two) business days** after the subject's study visit.

#### 3. OBJECTIVES

| Primary Objectives | Corresponding Primary Endpoint |
|---|---|
| <b>Phase 1b:</b> To determine the safety and | |
| tolerability of neoadjuvant talimogene | Incidence of DLTs |
| laherparepvec in combination with | |
| preoperative EBRT as assessed by incidence | |
| of dose-limiting toxicities (DLT) in subjects | |
| with locally advanced high grade soft tissue | |

| sarcomas. | |
|---|---|
| Phase 2: To estimate the efficacy of neoadjuvant talimogene laherparepvec and radiotherapy as assessed by the pathological complete response rates (pCR) in subjects with histologically confirmed diagnosis of locally advanced STS that is unresectable with clear wide margins, for which preoperative radiotherapy is considered appropriate. | pCR rate - the proportion of subjects with pathologic tumor necrosis ≥90% |
| Secondary Objectives | Corresponding Secondary Endpoint |
| Further assess the safety of talimogene laherparepvec given concurrently with preoperative external beam radiation in | Type, incidence, severity, and relatedness of AEs |
| sarcoma patients. | ORR – The proportion of subjects with a complete or partial response. |
| To estimate: | |
| Overall response rate (ORR) | TTP - Time from first day of study treatment |
| Time to progression (TTP) | to first documented disease progression |
| Overall survival (OS) | |
| | Overall survival – Time from first day of |
| | study treatment to death due to any cause. |

For this study, pCR will be defined as  $\geq$  90% tumor necrosis following concurrent radiation therapy and talimogene laherparepvec.

#### 4. PATIENT SELECTION

# 4.1 Eligibility Criteria

- **4.1.1** Subject has provided informed consent.
- **4.1.2** Histologically confirmed diagnosis of locally advanced STS that is unresectable with clear wide margins, for which preoperative radiotherapy is considered appropriate. **EXAMPLES:**

- Resectable stage IIB, III, and IV disease that are not suitable for surgically resection alone due to inability to achieve clear margins.
- Including metastatic (stage IV) disease for which radiotherapy and surgical resection are indicated.
- Except certain histologic subtypes: GIST, Desmoid, Ewing sarcoma, Kaposi sarcoma, bone sarcomas and myxoid liposarcomas (Grade 1)
- **4.1.3** Previous treatment: prior systemic anti-cancer treatment consisting of chemotherapy, immunotherapy, or targeted therapy are allowed provided therapy completed at least 1 year prior to enrollment.
  - No prior Talimogene laherparepvec or tumor vaccines allowed.
  - No prior radiation to the same tumor bed allowed.
- **4.1.4** Age  $\ge 18$  years.
- **4.1.5** Both men and women of all races and ethnic groups are eligible for this trial.
- **4.1.6** ECOG performance status  $\leq 1$ .
- **4.1.7** Patient must have measurable disease:
  - Tumor size at least  $\geq$  5 cm in the longest diameter as measured by CT scan or MRI for which radiation is feasible.
- **4.1.7.1** Patient must have injectable disease (direct injection or ultrasound guided).
- 4.2 Exclusion Criteria
- **4.2.1** Certain histologic subtypes: GIST, Desmoid, Ewing sarcoma, Kaposi sarcoma, bone sarcomas and low grade myxoid liposarcomas (Grade 1)
- **4.2.2** History or evidence of sarcoma associated with immunodeficiency states (e.g.: Hereditary immune deficiency, HIV, organ transplant or leukemia).
- **4.2.3** Subjects with retroperitoneal and visceral sarcoma.
- **4.2.4** History or evidence of gastrointestinal inflammatory bowel disease (ulcerative colitis or Crohn's disease) or other symptomatic autoimmune disease including, inflammatory bowel disease, or history of any poorly controlled or severe systemic autoimmune disease (i.e., rheumatoid arthritis, systemic lupus erythematosus, scleroderma, type I diabetes, or autoimmune vasculitis).
- **4.2.5** History of other malignancy within the past 3 years except treated with curative intent and no known active disease present and has not received chemotherapy for  $\geq 1$  year before enrollment/randomization and low risk for recurrence.


- **4.2.6** History of prior or current autoimmune disease.
- **4.2.7** History of prior or current splenectomy or splenic irradiation.
- **4.2.8** Active herpetic skin lesions
- **4.2.9** Require intermittent or chronic treatment with an anti-herpetic drug (e.g., acyclovir), other than intermittent topical use.
- **4.2.10** Any non-oncology vaccine therapies used for the prevention of infectious disease within 28 days prior to enrollment and during treatment period.
- **4.2.11** Concomitant treatment with therapeutic anticoagulants such as warfarin. Patients on therapeutic low molecular weight heparin may be allowed provided the dose can be safely held as per the treating investigator on the morning of scheduled intratumoral injection and can be resumed 12 hours after the procedure.
- **4.2.12** Known human immunodeficiency virus (HIV) disease (requires negative test for clinically suspected HIV infection).
- **4.2.13** Acute or chronic hepatitis B or hepatitis C infection (requires negative test forclinically suspected hepatitis B or hepatitis C infection).
  - Evidence of hepatitis B -
    - 1. Positive HBV surface antigen (indicative for chronic hepatitis B or recent acute hepatitis B).
    - 2. Negative HBV surface antigen but positive HBV total core antibody (indicative for resolved hepatitis B infection or occult hepatitis B) and detectable copies of HBV DNA by PCR (detectable HBV DNA copies suggest occult hepatitis B).
  - Evidence of hepatitis C -
    - 1. Positive HCV antibody and positive HCV RNA by PCR (undetectable RNA copies suggest past and resolved hepatitis C infection).
- **4.2.14** Female subjects who are pregnant or breast-feeding, or planning to become pregnant during study treatment and through 3 months after the last dose of study treatment.
- **4.2.15** Female subjects of childbearing potential or male subjects who are unwilling to use 2 highly effective methods of contraception during study treatment and through 3 months after the last dose of study treatment. See Section 7.5 for more details.
- **4.2.16** Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(s).
- **4.2.17** Other investigational procedures while participating in this study that could affect the primary objective of the study as determined by the PI are excluded.


- **4.2.18** Subject previously has entered this study.
- **4.2.19** Patients who are receiving any other investigational agents.
- **4.2.20** Evidence of CNS metastases.
- **4.2.21** History of allergic reactions attributed to compounds of similar chemical or biologic composition to talimogene laherparepvec.
- **4.2.22** Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
- **4.2.23** Patients on or requiring immunosuppressive therapies.
- **4.2.24** Any of the following laboratory abnormalities:
  - Hemoglobin < 9.0 g/dL
  - Absolute neutrophil count (ANC) < 1500 per mm<sup>3</sup>
  - Platelet count < 100,000 per mm<sup>3</sup>
  - Total bilirubin > 1.5 × ULN
  - Aspartate aminotransferase (AST) or alanine aminotransferase (ALT)  $> 2.5 \times ULN$
  - Alkaline phosphatase  $> 2.5 \times ULN$
  - PT (or INR) and PTT (or aPTT)  $> 1.5 \times ULN$
  - Creatinine  $> 2.0 \times ULN$

#### 5. TREATMENT PLAN AND STUDY SCHEMA

#### 5.1 Study Design

This is a single-arm open-label phase Ib and phase II clinical study assessing the safety and relative efficacy of concurrent talimogene laherparepvec in combination with radiotherapy in patients with soft tissue sarcomas. Patients will be treated with neoadjuvant radiation and weekly intratumoral injections of talimogene laherparepvec. Weekly injections of talimogene laherparepvec will be continued until surgery. Surgery will be performed 4-6 weeks from the end of radiation therapy to allow for resolution of acute toxicities per current standard of care.

#### Phase 1b:

The phase Ib portion of this study is to ensure the safety and tolerability of talimogene laherparepvec in combination with EBRT as assessed by incidence of dose-limiting toxicities (DLT). Although this combination has been shown to be safe and well tolerated in several other tumor types including melanoma and head & neck cancers, this combination has not been studied in sarcoma patients. EBRT will be given at the standard dose for resectable soft tissue

sarcomas according to the NCCN sarcoma guidelines.<sup>2</sup> Patients will receive 50 Gy over 5 weeks, during which time they will be receiving weekly injections of talimogene laherparepvec. Weekly injections of talimogene laherparepvec will be continued until surgery 4-6 weeks later. Surgery will be performed 4-6 weeks from the end of radiation to allow for adequate tissue healing and resolution of acute toxicities.

Talimogene laherparepvec will be dosed at an initial dose of up to 4.0 mL of 10<sup>6</sup> PFU/mL on day 1 of week 1, followed by the target dose of up to 8.0 mL of 10<sup>8</sup> PFU/mL (Dose 0) three weeks later on day 1 of week 4, and dosed weekly until surgery. Initially 3 patients will be entered at the Dose 0 (following initial dose of up to 4.0 mL of 10<sup>6</sup> PFU/mL on day 1 of week 1) for talimogene laherparepvec and be monitored at this weekly dose through 4 injections, when safety issues will be addressed. Data from safety analysis will be reviewed with Amgen Medical and Safety team. If none or one of the 3 patients shows a DLT, three more patients will be entered into the study at this dose and be monitored at this weekly dose through 4 injections. If none or one of these 6 patients shows a DLT, this is the dose that will be used for the phase II relative efficacy assessment. Otherwise, talimogene laherparepvec dose will be deescalated and dose -1 will be explored as outlined below in Table 1. For this protocol DLT will be defined as an attributed adverse event (definite, probable or possible) that meets the criteria in Section 6.2.

#### Phase 2:

The phase 2 part of the study will provide an estimate of the relative treatment effect of talimogene laherparepvec in combination with preoperative EBRT in subjects with histologically confirmed diagnosis of locally advanced STS that is unresectable with clear wide margins, for which preoperative radiotherapy is considered appropriate, as measured by pathological response rates. Twenty- eight (28) patients will be enrolled into the phase 2 portion of this protocol.

As above, patients will receive the first dose of talimogene laherparepvec 4.0 mL of 10<sup>6</sup> PFU/mL on day 1 of week 1, and followed three weeks later by weekly injections at Dose 0. Weekly injections of talimogene laherparepvec will be continued until surgery. The EBRT will be given at the standard dose for resectable soft tissue sarcomas according to the NCCN sarcoma guidelines.<sup>2</sup> Patients will receive preoperative radiation at a dose of 50 Gy over 5 weeks starting around week 4, and continued concurrently with weekly injections of talimogene laherparepvec. Subjects should be followed by clinic visit every 12 weeks for approximately 24 months after the end of the treatment phase, at which time the initial survival data and disease recurrence will be assessed. Subjects will be followed for an additional 3 years for survival and disease recurrence after that according to the standard-of-care. Please see study calendar in Section 10.

#### **Study Timeline Schema:**



First dose of TVEC

Complete XRT

Complete TVEC→ MRI of tumor→ then Surgery

#### Phase 1b schema:



#### Phase 2 schema:



#### **Talimogene Laherparepvec Dose Levels:**

Dose  $0 = \text{talimogene laherparepvec up to } 8.0 \text{ mL of } 10^8 \text{ PFU/mL dosed weekly}$ Dose  $-1 = \text{talimogene laherparepvec up to } 8.0 \text{ mL of } 10^8 \text{ PFU/mL dosed every } 2 \text{ weeks.}$ 

• Initial dose for all = talimogene laherparepvec up to 4.0 mL of 10<sup>6</sup> PFU/mL

#### Rationale for Talimogene Laherparepvec Dosing

Multiple studies have documented the efficacy and safety of talimogene laherparepvec in melanoma and head and neck cancer patients. 24-26 In a phase I study to evaluate the safety, biodistribution, and biological activity of differing dose levels of talimogene laherparepvec in patients with advanced solid tumors. Hu et al identified that subjects who are seronegative for HSV-1 more commonly developed febrile flu-like symptoms and erythematous skin rashes at higher initial doses of talimogene laherparepvec (10<sup>7</sup> and 10<sup>8</sup> PFU/mL) compared to a decreased initial dose of 10<sup>6</sup> PFU/mL.<sup>27</sup> Additionally, in a phase I/II upward-titration study to assess the safety and biological activity of three dose levels of talimogene laherparepvec (all initial doses were 10<sup>6</sup> PFU/mL, followed by subsequent doses of 10<sup>6</sup>, 10<sup>7</sup> or 10<sup>8</sup> PFU/mL) a greater mean decrease in tumor size was observed in patients receiving subsequent doses of 10<sup>7</sup> PFU/mL or higher compared to those administered only 10<sup>6</sup> PFU/mL for all doses. The study also reported that none of the injected tumors in the lowest dose cohort (10<sup>6</sup> PFU/mL) had resolved by the end of the treatment period, whereas 36.5% (12/32) of measurable tumors resolved (i.e., were no longer detectable) at the higher dose levels, suggesting that talimogene laherparepvec has a doserelated effect on tumor necrosis.<sup>26</sup> For this study all subjects will be treated with an initial dose of talimogene laherparepvec 10<sup>6</sup> PFU/mL, followed by 10<sup>8</sup> PFU/mL for all subsequent doses in accordance with the currently approved maximum tolerated dosing per the above phase I studies. A Phase 1b/2 trial in patients with advanced soft tissue sarcomas of the trunk and extremities was conducted at University of Iowa. As per the safety results presented there were no dose limiting toxicities noted at doses of 4 mL of 10<sup>8</sup>PFU/mL. One of the possibilities for failure to reach the primary endpoint was the lower amount of drug injected relative to the size of sarcomas. Hence a trial amendment with higher injectable dose of the drug is being proposed.

# 5.2 Study Agent Administration: Talimogene Laherparepvec

# **5.2.1** Talimogene Laherparepvec Dose Levels:

- Initial dose for all = talimogene laherparepvec up to 4.0 mL of 10<sup>6</sup> PFU/mL
- Dose  $0 = \text{talimogene laherparepvec up to } 8.0 \text{ mL of } 10^8 \text{ PFU/mL dosed weekly}$
- Dose -1 = talimogene laherparepvec up to 8.0 mL of 10<sup>8</sup> PFU/mL dosed every 2 weeks.

#### Dosing Schedule:

Patients will be treated with 50 Gy over 5 weeks and concurrent weekly injections of talimogene laherparepvec. Weekly injections of talimogene laherparepvec will be continued until surgery, about 4-6 weeks later.

#### Dosing Information:

Talimogene laherparepvec will be only administered by intratumoral injection into soft tissue tumors with or without image ultrasound guidance. Talimogene laherparepvec must not be administered into visceral organ metastases.

The initial dose of talimogene laherparepvec is up to 4.0 mL of  $10^6$  PFU/mL. Subsequent doses of talimogene laherparepvec are up to 8.0 mL of  $10^8$  PFU/mL. The maximum volume of talimogene laherparepvec administered at any dose is 8.0 mL for any individual lesion. The maximum dose in any one treatment is 8.0 mL. Investigators are encouraged to use the

maximum amount whenever lesions allow. In response to severe AEs, dose delays and dose descalations may be employed, but dose volume reduction for AEs is not allowed – see Section 6. However if in the course of administration of talimogene laherparepvec the subject cannot tolerate the full dose due to an injection-related AE such as pain, the total volume given should be recorded, and the reason for intolerance should be documented as an AE.

Treatment will be administered on an outpatient basis. Reported adverse events and potential risks are described in Section 7. Appropriate dose modifications are described in Section 6. No investigational or commercial agents or therapies other than those described below may be administered with the intent to treat the patient's malignancy.

#### **5.2.2** Lesion site preparation

- Talimogene laherparepvec is only to be administered by intralesional injection into soft tissue tumors with or without image ultrasound guidance. Talimogene laherparepvec must not be administered into visceral organ metastases.
- The injection site may be pre-treated with a topical anesthetic agent or an injectable local anesthetic; however, a local anesthetic must not be injected directly into the lesion.
- Swab the lesion and surrounding areas with alcohol, allow to dry.

### 5.2.3 Lesion injection

- All personnel handling talimogene laherparepvec or material contaminated with talimogene laherparepvec must observe safety precautions (e.g., wear a laboratory coat, safety glasses and gloves).
- Inject talimogene laherparepvec intralesionally:
  - a) A single point of insertion is recommended; multiple insertion points may be used if the tumor is larger than the radial reach of the needle.
  - b) Talimogene laherparepvec should be injected along multiple different tracks within the lesion in order to obtain as wide dispersion as possible.
  - c) Distribute talimogene laherparepvec within the lesion through the insertion point using the radial reach of the needle in different directions to evenly distribute.



- Avoid premature extraction of needle.
- After dosing, the injection site should be swabbed with alcohol and pressure should be applied with gauze for several seconds after injection.
- The injection site should be covered with an absorbent pad and dry occlusive dressing.
- Dispose materials used during injection (e.g., gloves, needles, gauze) in accordance with local/regional and institutional requirements for biohazardous waste.

#### 5.2.4 Radiation Therapy

External beam radiation therapy will be given at the standard dose for resectable soft tissue sarcomas according to the NCCN sarcoma guidelines.<sup>2</sup> Patients will receive 50 Gy over 5 weeks, during which time they will be receiving weekly injections of talimogene laherparepvec. Weekly injections of talimogene laherparepvec will be continued until surgery 4-6 weeks later. Surgery will be performed 4-6 weeks from the end of radiation to allow for adequate tissue healing and resolution of acute toxicities.

Radiation therapy for this protocol is as per currently used standard pre-operative radiation therapy at the University of Iowa even for non-protocol patients.

Selected guidelines from previously conducted Radiation Therapy Oncology Groups (RTOG) studies are briefly summarized for this protocol.

#### **Preoperative Radiation therapy (3D-CRT or IMRT)**

Either 3D conformal radiotherapy or intensity modulated radiation therapy may be utilized for adequate tumor coverage and to meet the dose constraints for critical normal structures.

#### Radiation treatment planning scans and immobilization:

CT scans with patient in a stable and comfortable position will be used for planning. MRI scans are optional and may be used for co-registration with CT for tumor localization as needed. VacLoc or other immobilization devices can be used for immobilization.

### Target volumes and treatment field:

Gross Target Volume (GTV): Outline of the tumor as seen on CT or CT/MRI fusion. Clinical Target Volume (CTV): CTV = GTV plus 4 cm margins in the proximal and distal directions. However the margin can be reduced if it extends beyond the compartment, the field can be shortened to include the end of a compartment. The radial margin from the lesion should be 1 cm. It can be reduced in areas confined by the fascial barrier or bone or skin surface. Planning Target Volume (PTV): Include CTV and error of setup and organ motion. Typically PTV includes CTV plus 1 cm in all dimensions. Final PTV is usually GTV + 5 cm longitudinal and 2 cm radial, except where restricted by the compartment end, fascia, bone or skin surface. Use of bolus on the skin surfaces is optional as needed. Where applicable, biopsy scars should be bolused with appropriate thickness specific to the energy of the photon beam.

#### **Dose Specifications:**

A dose of 50 Gy in 25 daily fractions will be prescribed to the planning target volume (PTV) using linear accelerator and megavoltage photon beams with energies of 6MV or greater. Prescribed dose should cover > 90% of the PTV. More than 95% of the PTV should receive > 95% of the prescribed dose. No more than 20% of the PTV will receive  $\ge 110\%$  prescription dose.

#### **Precautions and Dose Constraints for critical structures:**

Radiation dose to normal tissues should be kept within the accepted normal tissue tolerances. Every effort should be made to:

- a) Avoid treating the full circumference of an extremity;
- b) Avoid treating anus, urogenital tract, perineum and genitalia; if the tumor is close to these structures, typically less than 50% volume of the anus and vulva should receive 30 Gy; less than


50% volume of the testis should receive 3 Gy, if the patient prefers to reserve fertility;

- c) Avoid treating the lung, through use of appropriate shielding and treatment planning; less than 20% of the lungs should receive 20 Gy (V20);
- d) Avoid dose maximums in areas where surgical scars will be placed; this may require reviewing treatment plans with the surgeon;
- e) If possible, avoid treating skin over areas commonly traumatized to full dose (e.g., theelbow, knee, shin, femoral neck).
- f) If possible, less than 50% of any joints (including shoulder, elbow and knee) should receive 50 Gy.
- g) Less than 50% of kidney volumes should receive 18 Gy.
- h) No more than 50% of normal weight-bearing bone within the radiation field should receive 50 Gy except when the tumor invades the bone or when there is circumferential involvement of the tumor more than a quarter of the bone or when the bone will be resected in a subsequent surgical resection after radiation.

For any other normal tissue structures, no radiation dose more than the established TD5/5 limit should be given.

#### **Image Guidance and Verification Devices**

Portal films or conebeam CT images should be used for target localization and alignment. Daily conebeam CT will be preferred and dose from daily conebeam should be included in the final dosimetry.

## **Postoperative Radiotherapy Boost**

External Beam or Brachytherapy boost can be given at the discretion of the radiation oncologist, to the positive tumor margin (residual tumor) only plus a margin of 1 cm within 2 weeks following surgery or after adequate wound healing has occurred.

The target volume for postoperative radiotherapy will be the residual tumor bed as defined by the surgical and pathological findings.

#### **External Beam Radiotherapy**

Postoperative external beam boost dose is 16 Gy in 8 fractions (once a day).

# **Brachytherapy**

High-dose-rate (HDR) brachytherapy as a boost to the positive tumor margin can be used as an alternate to external beam radiotherapy. Brachytherapy catheters are placed at an interval of 0.5 -1.0 cm on the residual tumor bed (positive margin) plus a margin of 1 cm during surgery. Skin surface dose should be kept below 50% of the prescription dose unless positive margins occur in cutaneous or subcutaneous tissues. It is not necessary to include the entire surgical bed, drain sites and wound. Brachytherapy should not start until day 5 after the surgery (day 0) and must be completed within 2 weeks following surgery.

For HDR brachytherapy, 4 fractions of 3.4 Gy are delivered b.i.d, with an interval of at least 6 hours between fractions.

#### **Radiation Therapy Adverse Events**


Acute: Wound complications of any grade are expected to develop in about one third of patients. Other common radiation adverse events include: fatigue, regional alopecia, diarrhea, skin erythema and desquamation within the treatment fields, and reduction in blood counts. Long-term: Common long-term treatment adverse events include: lymphedema of the extremity receiving radiation and surgery, subcutaneous fibrosis, and joint stiffness. Much less common radiation adverse events include bowel injury, osteoradionecrosis, and bony fracture in the radiation field. There also is a risk of secondary malignancy occurring in the irradiated field.

#### 5.3 General Concomitant Medication and Supportive Care Guidelines

Patients should receive full supportive care, including transfusions of blood and blood products, antibiotics, antiemetics, etc., when appropriate. The reason(s) for treatment, dosage, and the dates of treatment should be recorded.

All other protocol-required therapies including, topical anesthetic or an injectable local anesthetic medications used for pretreatment of the talimogene injection site and oral or systemic treatments required for management of immune-mediated AEs that are to be obtained commercially.

Throughout the study, investigators may prescribe any concomitant medications or treatments deemed necessary to provide adequate supportive care. All prescription and nonprescription concomitant medication administered up to 28 days prior to enrollment, on an ongoing basis at enrollment, as well as changes in such concomitant medication, and any new concomitant medication taken while the subject is on study, should be recorded up to 30 days after the last dose of talimogene laherparepvec.

# 5.4 Duration of Therapy

Concurrent immunoradiotherapy with a total of 50 Gy of radiation and weekly talimogene laherparepvec intratumoral injections will be given over 5 weeks. Then, weekly intratumoral injections of talimogene laherparepvec will be continued until surgery is performed around 4-6 weeks later. In the absence of treatment delays due to adverse event(s), treatment may continue until surgical resection of the tumor, or until one of the following criteria applies:

- Intercurrent illness that prevents further administration of treatment,
- Unacceptable adverse event(s),
- Patient decides to withdraw from the study, or
- General or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator.

#### 5.5 **Duration of Follow Up**


#### Safety Follow up Visit

Upon permanent discontinuation from the study treatment for any reason, the following procedures will be performed approximately 30 (+7) days after the last dose of Talimogene Laherparepvec:

- Recording of concomitant medications and AE/SAE(s)
- Physical examination including weight, vital signs and ECOG performance status assessment
- Local laboratory tests including the following:
  - Hematology panel
  - Chemistry panel
  - o Serum or urine pregnancy test for female subjects of childbearing potential

## Long-term Follow up

Following the end of treatment, subjects will be followed according to standard of care (approximately every 12 -16 weeks +/- 2 weeks), as per NCCN guidelines and at the discretion of the treating physician, at which time disease recurrence and survival status will be assessed for up to 5 years. Data for disease recurrence and survival status only will be collected per chart review, phone call or email.

#### End of Study

The end of study for each subject is defined as the date the subject withdraws full consent from the study, completes the safety follow-up visit or the long-term survival follow-up whichever is later, or death.

#### 5.6 Criteria for Removal from Study

Talimogene laherparepvec is to be permanently discontinued for subjects meeting any of the following criteria:

- The subject, for any reason, requires treatment with another anticancer therapeutic agent for treatment of the study disease (other than the exceptions noted in protocol, if applicable). In this case, discontinuation from the treatment occurs immediately upon introduction of the new agent.
- Clinical relevant disease progression as defined in the study protocol.
- Immune-mediated adverse events have been observed in subjects receiving talimogene laherparepvec. These have included pauci-immune glomerulonephritis, vasculitis, and pneumonitis; however, immune-mediated adverse events can potentially involve any organ system. Permanently discontinue talimogene laherparepvec if dosing is delayed by more than 4 weeks due to a Grade 2 or greater immune-mediated adverse event (with the exception of vitiligo), allergic reactions, or urticaria attributed to talimogene laherparepvec.
- Plasmacytoma has been observed with the administration of talimogene laherparepvec.
   Permanently discontinue talimogene laherparepvec if development of a plasmacytoma is observed.


- Any talimogene laherparepvec-related non-hematologic or hematologic toxicities Grade 3 or greater that, in the opinion of the investigator, would require a dose delay of greater than 4 weeks or discontinuation of therapy.
- A female subject becomes pregnant or fails to use 2 highly effective methods of contraception (for those subjects who are able to conceive).
- A female subject breast feeds while on study treatment.
- A male subject fails to use a highly effective method of contraception as described in Section 7.5.
- Intercurrent medical illness that, in the judgment of the investigator, would make continued treatment with talimogene laherparepvec dangerous for the subject.

#### 6. DOSING DELAYS/DOSE MODIFICATIONS

#### 6.1 Dose Delays

If talimogene laherparepvec treatment was delayed due to adverse events or other reasons by > 1 week, that dose will be deemed to have been missed and the subject will proceed to the next scheduled treatment visit.

If dose-limiting toxicities occur, talimogene laherparepvec administration should be delayed until the DLT has resolved to at least CTCAE version 4.0 Grade 1 (see Appendix E). Dosing of talimogene laherparepvec could also be delayed for active herpetic cutaneous or mucosal lesions, herpes labialis, or active dermatoses in the region of the injected tumors. Talimogene laherparepvec should be discontinued for subjects with evidence of systemic herpetic infection, herpetic keratitis, encephalitis, or evidence of other disseminated herpetic infection or any herpetic infection requiring treatment with acyclovir or a similar agent.

If talimogene laherparepvec dosing is delayed by more than 4 weeks due to the occurrence of DLT or adverse events that are related to talimogene laherparepvec, then treatment should be discontinued. If talimogene laherparepvec dosing is delayed by more than 4 weeks for reasons other than treatment-related toxicity, the case must be reviewed by the sponsor of the investigator sponsor study (ISS) to determine if the subject can resume talimogene laherparepvec therapy.

If the subject requires corticosteroid dosing of > 10 mg prednisone daily (or equivalent) and/or other immunosuppressive medication for related toxicities, talimogene laherparepvec dosing must be held until the corticosteroid dose has decreased to < 10 mg prednisone daily (or equivalent) and the administration of the other immunosuppressive medication has discontinued.

#### **6.2** Dose Limiting Toxicities

Definitions of dose-limiting toxicity:


Toxicity will be evaluated according to CTCAE version 4.0. DLT will be defined as any of the following talimogene laherparepvec-related toxicity or related to the combination of talimogene laherparepvec and radiation therapy during treatment and through week 8:

- Grade 3 or greater immune-mediated adverse events
- Grade 3 or greater allergic reactions.
- Any grade plasmacytoma
- Any other unexpected grade 3 or greater hematologic or non-hematologic toxicity, with the exceptions of:
  - Any grade of alopecia.
  - Expected radiation related skin toxicity of any grade.
  - Grade 3 arthralgia or myalgia.
  - Brief (< 1 week) grade 3 fatigue.
  - Grade 3 fever.
  - Grade 3 diarrhea or vomiting responding to supportive case.

Of note, unless an alternative etiology has been identified, signs and symptoms of any disease process described above as a DLT should be considered immune-mediated.

If unexpected DLT occurs, talimogene laherparepvec administration should be delayed until the DLT has resolved to at least CTCAE version 4.0 grade 1. If dosing is delayed by more than 4 weeks due to the occurrence of unexpected adverse event that is considered related to talimogene laherparepvec, then the subject should be taken off treatment.

### **6.3** Dose Reductions

Dose reductions with regards to changes in the concentrations of talimogene laherparepvec are not permitted.

- Patients may require a reduction in the volume injected due to a disease response as outlined in Section 5.1.
- Additionally, subjects who miss two consecutive doses of talimogene laherparepvec due to a DLT should be reduced to a biweekly dosing (dose -1 as in section 5.1).

#### 7. ADVERSE EVENTS: LIST AND REPORTING REQUIREMENTS

Adverse event (AE) monitoring and reporting is a routine part of every clinical trial. The following list of AEs (Section 7.1) and the characteristics of an observed AE (Section 7.2) will determine whether the event requires expedited reporting **in addition** to routine reporting.

Information regarding the occurrence of adverse events will be collected from the time the subject signs the informed consent form and throughout their participation in the study, including a period of 30 days after the last dose of study drug (data on serious adverse events (SAEs) will be collected until resolution of the event unless otherwise noted). Serious adverse events occurring outside the 30-day follow-up period, which are assessed as related to study drug, should be reported to Amgen, along with any SAE that the investigator feels should be reported.

#### 7.1 Adverse Event Definitions

An **adverse event** (AE) is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An adverse event can be any unfavorable and unintended sign including clinically significant abnormal laboratory finding, symptom, or disease temporally associated with the use of the drug, without any judgment about causality. This includes any newly occurring event or previous condition that has increased in severity or frequency since the administration of drug.

Following surgical resection of the tumor, non-serious adverse events consistent with an expected post-operative course will not be reported unless attributable to the study drug and/or meet the seriousness criteria.

An adverse event is considered a **serious adverse event** (SAE) if it results in any of the following outcomes:

- 1) Results in death
- 2) Is a life-threatening event (ie, its occurrence places the patient or subject at immediate risk of death)
- 3) Requires inpatient hospitalization or prolongation of existing hospitalization for  $\geq$  24 hours
- 4) Results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- 5) Is a congenital anomaly/birth defect
- 6) Is an important medical event that may not result in death, be life threatening, or require hospitalization but may be considered serious when, based upon medical judgment, may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

#### **Suspected Adverse Reaction**

Suspected adverse reaction means any adverse event for which there is a reasonable possibility that the drug caused the adverse event. For the purposes of IND safety reporting, 'reasonable possibility' means there is evidence to suggest a causal relationship between the drug and the adverse event. A suspected adverse reaction implies a lesser degree of certainty about causality than adverse reaction, which means any adverse event caused by a drug.

# **Unexpected Adverse Events**

An adverse event is considered "unexpected" if it is not listed in the table of expectedness within the Investigator Brochure or is not listed at the specificity or severity that has been observed; or, if an Investigator Brochure is not required or available, is not consistent with the risk information described in the general investigational plan or elsewhere in the current application.

When talimogene laherparepvec is administered in combination with 1 or more approved antineoplastic agents, the expectedness determination should take into account the labeling of each specific marketed drug taken in combination based upon reference documents which will be included or referenced in the clinical study protocol. The labeled events should, in general, be


considered expected for at least one of the drugs in the combination. The contribution of talimogene laherparepvec to the severity or frequency of the events is currently unknown. See Section 1.2.2 for adverse drug reactions that could be reasonably assumed to be associated with talimogene laherparepvec.

#### 7.2 Adverse Event Characteristics

CTCAE term (AE description) and grade: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version4.0 (Appendix E) will be utilized for AE reporting. If specific grading is not available in the CTCAE for a particular AE's severity/intensity, the Investigator is to revert to the general definitions of Grade 1 through 5 and use his/her best medical judgment. The 5 general grades are: Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life-threatening or disabling, Grade 5 = death related to AE.

#### **Attribution** of the AE:

Investigators are required to assess whether there is a reasonable possibility that talimogene laherparepvec caused or contributed to the adverse event. The following general guidance may be used.

- Definite The AE *is clearly related* to the study treatment.
- Probable The AE *is likely related* to the study treatment.
- Possible The AE *may be related* to the study treatment.
- Unlikely The AE *is doubtfully related* to the study treatment.
- Unrelated The AE *is clearly NOT related* to the study treatment.

# 7.3 Comprehensive Adverse Events and Potential Risks List (CAEPR)

All necessary supportive care shall be available to subjects. Additional treatment modifications should be considered depending upon the subject's clinical situation. Talimogene laherparepvec treatment should be continued based on the potential risk/benefit assessment of the subject.

#### 7.3.1 Important Identified Risks

#### Accidental Exposure of Healthcare Providers (HCP) to Talimogene Laherparepvec

A needle stick injury, spill, or splash back during administration may result in accidental exposure of HCPs to talimogene laherparepvec. The ICP34.5 gene deletion is intended to allow only tumor selective replication and limited or no viral replication in normal tissues. However, talimogene laherparepvec injection can result in signs or symptoms of primary infection at the site of exposure. A few reports of accidental exposure in study personnel have been received. In one of the cases, the exposed physician developed clinical signs/symptoms of a herpetic whitlow-like lesion at the site of the accidental needle stick injury that resolved without sequelae. An initial antibody assay was positive for an HSV-type virus. A confirmatory PCR assay was conducted 10 days after the accidental exposure and was positive for a virus with the ICP47 deletion, indicating that the virus was most likely talimogene laherparepvec. None of the other exposed individuals reported signs or symptoms of infection. In some cases oral acyclovir or valacyclovir was administered.

#### **Cellulitis at Site of Injection**

Intralesional administration of talimogene laherparepvec by injection has been associated with cellulitis at the injection site. In some cases, a local inflammatory reaction with localized tumor necrosis developed, and in other cases, a bacterial infection developed. In the pivotal clinical study, the subject incidence of adverse events in the bacterial cellulitis category was 6.2% (n = 18) in the talimogene laherparepvec group and 1.6% (n = 2) in the GM-CSF group. The most frequently reported preferred term was cellulitis (5.8% in the talimogene laherparepvec group and 1.6% in the GM-CSF group). Seven subjects (2.4%) in the talimogene laherparepvec group and 1 subject (0.8%) in the GM-CSF group experienced serious adverse events of cellulitis. Fever, elevated white blood cell count, bacteremia or sepsis, and hospitalization for intravenous antibiotics were reported in 5 of the 7 cases in the talimogene laherparepvec group. Subjects should be monitored closely for cellulitis and injection site reactions.

#### Disseminated Herpetic Infection in Severely Immunocompromised Individuals

Patients with immunosuppression for any reason were excluded from clinical trials with talimogene laherparepvec. Disseminated herpetic infection in severely immunocompromised individuals is defined as an important identified risk based on the nonclinical data and literature described below. Evidence of lethal systemic viral infection was observed in 100% of severe combined immunodeficiency (SCID) mice (deficient in T and B cells) following intratumoral injection of talimogene laherparepvec in a mouse colon carcinoma xenograft model. Similar findings were observed in up to 20% of BALB/c nude mice (primarily deficient in T-cell function) following intratumoral injection of talimogene laherparepvec in Ewing's sarcoma and osteosarcoma xenograft models. Viral inclusion bodies and/or necrosis in enteric neurons in the gastrointestinal tract, adrenal gland, and skin were observed in both mouse strains; and in pancreatic Islet cells, eye, pineal gland, and brain of SCID mice. Lethality in 100% of animals following intracutaneous injection of wild-type HSV-1 in nude mice has been reported (Hayashida et al, 1982; Yamamoto et al, 1985). The data in talimogene laherparepvec treated SCID mice indicate that severe toxicity associated with disseminated viral infection may occur in patients who are severely immunosuppressed. The data in the BALB/c nude mice suggest the potential for toxicity due to talimogene laherparepvec in patients with less severe immunosuppression. Consistent with the general literature, these data indicate an important role of host defenses including T and B cells in the immune response to talimogene laherparepvec and HSV-1 viruses.

#### **Immune-mediated Adverse Events**

Based on review of adverse events suggestive of an immune-mediated etiology across melanoma studies, immune-mediated adverse events considered possibly related to talimogene laherparepvec were reported in 2% of subjects treated with talimogene laherparepvec, and included events of vasculitis, glomerulonephritis, acute renal failure, pneumonitis, and worsening psoriasis. Other contributory factors were identified in several of these cases, including pre-existing immune-mediated conditions, other concurrent medications, or intercurrent medical events.

#### Plasma Cell Dyscrasia (Plasmacytoma) at the Injection Site

A plasmacytoma was reported in 1 subject treated with talimogene laherparepyec in the pivotal


clinical study. A plasmacytoma developed in the area of the injected tumor on the scalp after 9 cycles of treatment with talimogene laherparepvec. Study treatment was permanently discontinued. On medical review, the event was determined likely to be a secondary plasmacytoma which developed at the injection site due to recruitment of plasma cells in response to the talimogene laherparepvec injections in a subject who had a pre-existing (smoldering) multiple myeloma.

Other important identified risks include obstructive airway disorder and deep vein thrombosis.

### 7.4 Important Potential Risks

# Symptomatic Talimogene Laherparepvec Infection in Non-tumor Tissue in Treated Patients

Talimogene laherparepvec is a modified HSV-1 virus, and is engineered to replicate selectively in tumor tissue. However, if infection by talimogene laherparepvec of non-tumor tissue in treated patients were to occur, this could lead to development of clinical signs or symptoms that would be anticipated to be similar to signs or symptoms of wild-type herpes virus infection.

In mouse tumor models, viral lysis/tissue injury was limited to tumors. No clinical or pathological evidence of symptomatic infection or injury to normal tissues was observed in nonclinical models dosed by repeated intratumoral, intravenous, or subcutaneous injection, including mice dosed with up to 107 PFU talimogene laherparepvec (~60-fold over the highest proposed clinical dose, on a PFU/kg basis) via weekly subcutaneous injection for up to 3 months.

No cases of confirmed infection of non-tumor tissue by talimogene laherparepvec in treated patients have been reported to date. In the pivotal clinical study, adverse events related to HSV infections were reported in 5.5% (n = 16) of subjects in the talimogene laherparepvec group and 1.6% (n = 2) in the GM-CSF group. Most of the cases were reported as oral herpes and 1 case each was reported as herpes simplex and herpetic keratitis in the talimogene laherparepvec group. The subject with herpetic keratitis had a history of this event prior to enrollment in the study. Whether the reported lesions were due to wild-type herpes or to talimogene laherparepvec could not be confirmed as viral testing was not performed.

# Transmission of Talimogene Laherparepvec from Patient to Close Contacts or HCPs Via Direct Contact with Injected Lesions or Body Fluids (eg, Blood or Urine) Resulting in Symptomatic Infection (Primary or Reactivation)

Proximity of close contacts and HCPs to lesions in treated patients in the absence of effective barriers may result in the unintentional exposure of these individuals to talimogene laherparepvec. Exposure may occur via direct contact with injected lesions or via contact with body fluids (eg, blood or urine). The likelihood of transfer of talimogene laherparepvec to a close contact or HCP increases if the contact has a break in the skin or mucous membranes. Signs or symptoms of infection would be anticipated to be similar to signs and symptoms of wild-type HSV infection.


Biodistribution by quantitative polymerase chain reaction (qPCR) testing in clinical studies indicated that low copy numbers of viral DNA were sporadically detected from 1 hour to 1 week after intratumoral injection in blood and urine in 30% of subjects across all studies. Where subsequent samples were available, no viral DNA was detected at 2 weeks after injection.

Shedding results showed that talimogene laherparepvec was detected on the surface of injected lesions for up to 2 weeks after injection in 8 of 72 (11%) subjects. Virus was not detected on the exterior surface of tumor dressings at any time point tested.

Biodistribution was evaluated after single and multiple dosing by intravenous, subcutaneous or intratumoral injection in mice. Doses from 1 x 105 to 1 x 107 PFU/mL were evaluated (0.6 to 60-fold higher compared to the maximum clinical dose). Across the studies, viral DNA was found most commonly at the site of injection regardless of administration route, which in the case of the tumor may reflect viral replication following intratumoral administration. Following intravenous administration of talimogene laherparepvec, viral DNA was detected in blood of 5 of 6 animals through 56 days of dosing. After intratumoral injection, talimogene laherparepvec DNA was detected by PCR in tumor, blood, in tissues associated with immune related viral clearance (lymph nodes, spleen), and tissues with high blood perfusion (heart, lung, liver). Viral DNA was found in the brain in 2 of 91 samples collected. Viral DNA was not detected in bone marrow, eyes, lachrymal glands, nasal mucosa or feces at any time point. Following intratumoral injection, viral DNA was cleared from the blood of most animals within 2 weeks postdose and in all animals by 6 weeks after the last dose. Following subcutaneous dosing, viral DNA was excreted in urine in 22% of animals within 24 hours postdose and all were negative at 4 weeks postdose.

# Symptomatic Herpetic Infection Due to Latency and Reactivation of Talimogene Laherparepvec or Wild-type HSV-1 in Patients

Infection of tumor or non-tumor tissue could potentially lead to the establishment of latency and subsequent reactivation of talimogene laherparepvec if the virus came into contact with axonal nerve terminals and was transported to neuronal cell bodies. The genetic modifications made to talimogene laherparepvec do not prevent the virus from entering latency or subsequently reactivating. However, HSV-1 strains deficient in the ICP34.5 gene are unable to replicate efficiently in non-tumor cells, including neurons, and are impaired for establishment and reactivation from latency when compared to wild-type HSV-1 (Chou et al, 1990; Perng et al, 1995; Perng et al, 1996, Robertson et al, 1992; Spivack et al, 1995). Thus, reactivated virus in nerve cells is expected to be less likely to lead to clinical signs or symptoms as compared to wild-type HSV-1.

Co-infection of neurons already harboring latent wild-type HSV-1 by talimogene laherparepvec could potentially stimulate the reactivation of latent wild-type HSV-1 in patients with prior infection. A febrile response associated with injection of talimogene laherparepvec might stimulate reactivation of wild-type HSV-1 in patients with prior exposure and latent HSV-1 infection.

Biodistribution studies in mice have detected low levels of talimogene laherparepvec in trigeminal ganglia (at levels 0.2-1.2% found in concurrent blood) through 28 days in 1 of 6


animals following high dose intravenous administration ( $0.6 \times 107$  PFU,  $\sim 36$ -fold over the highest proposed clinical dose). Talimogene laherparepvec was undetectable in trigeminal ganglia in mice after subcutaneous administration.

In a mouse model, talimogene laherparepvec was detected in the spinal dorsal root ganglia following injection into the foot. This suggests the virus had established latency in the nerve root innervating the site of injection. The virus was reactivated in ex vivo cell culture. The clinical applicability of these findings is not certain, as it is anticipated that host immunity will respond to protect the host from talimogene laherparepvec replication in non-tumor tissue in individuals with an intact immune system.

# Talimogene Laherparepvec-mediated Anti-GM-CSF Antibody Response

There is a theoretical concern that transgene-derived expression of GM-CSF could induce an immune response reactive with endogenous GM-CSF. Antibodies against GM-CSF have been detected sporadically in the general population (up to 9.6%) (Meager et al, 1999). Case reports of cryptococcal meningitis and pulmonary alveolar proteinosis have been reported in association with auto-antibodies to GM-CSF (Rosen et al, 2013). Auto antibodies to GM-CSF were demonstrated to reproduce the disease of pulmonary alveolar proteinosis in nonhuman primates (Trapnell et al, 2009). It is not known whether such phenomena could be expected with the limited exposure anticipated with transgene expression of GM-CSF from talimogene laherparepvec.

#### **Impaired Wound Healing at Site of Injection**

The local tissue response following repeated injections of a foreign protein can contribute to chronic inflammation, necrosis, and ulceration of tumor sites, and in the presence of other risk factors, delayed healing may result. In the pivotal clinical study, the incidence of adverse events in the impaired wound healing category was 5.5% (n = 16) in the talimogene laherparepvec group and 2.4% (n = 3) in the GM-CSF group. Wound complication, wound secretion, and wound infection were reported in  $\geq 1\%$  of subjects in the talimogene laherparepvec group. A serious adverse event of impaired healing was reported in an elderly subject following treatment with talimogene laherparepvec to a recurrent lower extremity melanoma lesion that resulted in a below the knee amputation 7 months after the last treatment. The subject had a history of peripheral vascular disease, prior radiation at the site of injection, and recurrent cellulitis in the area, all which were considered possible contributory factors. All subjects should be monitored very closely for impaired wound healing especially in the setting of concurrent use of radiation therapy.

Disseminated Herpetic Infection in Individuals with Deficiency in Cell-mediated Immunity Such as Human Immunodeficiency Virus (HIV)/Acquired Immunodeficiency Syndrome (AIDS), Lymphoma, or Leukemia, or Who Require High Dose Steroids or Other Immunosuppressive Treatments Such as Post Organ Transplant

Talimogene laherparepvec is a recombinant replication-competent HSV-1 type virus which is engineered to replicate selectively in tumor cells. Intratumoral injection of talimogene


laherparepvec was 100% lethal in SCID mice (SCID model) and in up to 20% of athymic mice (nude mouse model). Refer to the characterization of the important identified risk of "disseminated herpetic infection in severely immunocompromised individuals" for a description of results of nonclinical studies in SCID mice and BALB/c nude mice (Section 7.2.3).

The clinical relevance of these data to patients treated with talimogene laherparepvec is not clear. Wild-type HSV-1 infection in immunocompromised individuals is associated with dissemination of the virus and serious, life-threatening toxicity. Patients with immunosuppression were excluded from clinical trials with talimogene laherparepvec. The potential risk and potential benefits of treatment of patients with HIV/AIDS, leukemia, lymphoma, or patients who require treatment with chronic high dose steroids or other immunosuppressive agents such as those used in the post transplant setting should be considered prior to treatment. Talimogene laherparepvec is contraindicated in patients with severe immunodeficiency.

#### **Other Relevant Information**

Refer to the DCSI attached to this brochure as Appendix D for a description of current information related to adverse drug reactions, special warnings and precautions, contraindications, and risks for overdoses with talimogene laherparepvec.

# 7.5 PREGNANCY AND BREASTFEEDING

#### **Pregnancy**

No studies of the effects of talimogene laherparepvec on reproduction and development have been performed in humans. Talimogene laherparepvec should not be used during pregnancy.

#### **Females:**

Pregnant women and women planning to become pregnant should not receive talimogene laherparepvec. Women who can become pregnant must use 2 highly effective birth control methods (either by her alone or in combination with her male partner) during treatment with talimogene laherparepvec and for at least 3 months after the last tumor injection of talimogene laherparepvec. Highly effective methods of contraception include:

- Use of hormonal birth control methods: pills, shots, implants (placed under the skin by a health care provider) or patches (placed on the skin)
- Intrauterine devices (IUDs)
- Sexual activity with a male partner who has had a vasectomy (surgery to become sterile)
- Prior surgery to tie her fallopian tubes (surgery to become sterile)
- Condom or occlusive cap (diaphragm or cervical/vault caps) used with spermicide

If a woman becomes pregnant or suspects she is pregnant, she must tell her doctor immediately and treatment with talimogene laherparepvec will be stopped. The study doctor should notify Amgen of the pregnancy, discuss any follow-up with the subject, and ask for information on the pregnancy outcome.

#### Males:


The potential for talimogene laherparepvec to be transferred via semen and its effect on sperm are unknown. Males with partners of childbearing potential, must agree for the duration of the treatment with talimogene laherparepvec and continuing for 3 months after the last tumor injection of talimogene laherparepvec to practice a highly effective method of birth control, (either by him or his female partner). Highly effective methods of contraception include:

- Use of hormonal birth control methods: pills, shots, implants (placed under the skin by a health care provider) or patches (placed on the skin)
- Intrauterine devices (IUDs)
- Sexual activity with a male partner who has had a vasectomy (surgery to become sterile)
- Prior surgery to tie her fallopian tubes (surgery to become sterile)
- Condom or occlusive cap (diaphragm or cervical/vault caps) used with spermicide

If a pregnancy occurs, the study doctor must be notified. The study doctor should notify Amgen of the pregnancy, discuss any follow-up with the subject (and/or his partner), and ask for information on the pregnancy outcome. If the female partner is already pregnant when the male subject begins treatment with talimogene laherparepvec, he must refrain from any sort of sexual activity that could expose his partner or the unborn baby to talimogene laherparepvec through semen, or wear a condom during sexual activity while receiving treatment with talimogene laherparepvec and for at least 3 months after the last tumor injection of talimogene laherparepvec.

#### **Breast Feeding:**

Amgen has not tested whether talimogene laherparepvec is present in breast milk nor assessed the effects of talimogene laherparepvec in breast-fed infants. Therefore, babies should not be fed breast milk produced during treatment with talimogene laherparepvec or for an additional 3 months after the last tumor injection of talimogene laherparepvec.

#### 7.6 Other Relevant Information

Refer to Appendix D of this document and the DCSI in the latest version of the talimogene laherparepvec Investigator's Brochure for a description of current information related to contraindications and risks for overdoses with talimogene laherparepvec as well as information on the use of talimogene laherparepvec in special subject groups such as pregnant or breast feeding, pediatric, or geriatric populations.

#### 7.7 Expedited Adverse Event Reporting

## 7.7.1 Expedited Reporting Guidelines

Reporting to the HCCC DSMC per DSMP (Appendix E)

## **Reporting Requirements to AMGEN**

#### Safety Reporting to Amgen

The Sponsor/Investigator is responsible for compliance with expedited reporting requirements for serious, unexpected and related adverse events (SUSARs), for generation of SAE reports including narratives, and for periodic reporting to Amgen of SAEs as outlined in Table 2 and Table 3 below. Individual safety reports (Table 2) should be accompanied by the Fax Cover Form and sent to Amgen Global Safety, utilizing the fax of email information provided on the cover page. Aggregate safety reporting (Table 3) including listings, tabulations and summary reports should be scanned and accompanied by the Fax Cover Form and sent to Amgen NASCR, utilizing the email information provided on the cover page.

In addition to the requirements outlined in Table 2 and 3, Sponsor/Investigators are required to report **direct exposures** to talimogene laherparepvec (e.g., needle stick, splash back) of herpetic illness and **all suspected herpetic events** (refer to Section 'Accidental Exposures to Talimogene Laherparepvec and Herpetic Events').

**Table 2. Reporting Requirements for Interventional Studies** 

| Safety Data | Timeframe for Submission to Amgen |
|---|---|
| Suspected Unexpected Serious Adverse Reaction | Individual reports sent to Amgen at time of |
| (SUSARs) | expedited reporting to IRB and/or FDA. |
| Serious Adverse Events (SAEs) (related) | Individual reports sent to Amgen at time of |
| | expedited reporting to IRB and/or FDA. |
| Pregnancy/Lactation | Individual reports sent within 10 days of |
| | Sponsor/Investigator awareness. |

Individual reports should be faxed to 1-888-814-8653 or scanned and sent via email to <u>svc-ags-in-us-</u>@amgen.com.

**Table 3. Aggregate Reports:** 

| Safety Data | Timeframe for Submission to Amgen |
|---|---|
| Adverse events (all serious and non-serious | Line listing and summary tabulation of all adverse |
| adverse events, regardless of relatedness) | events sent annually AND at end of study |
| US IND Annual Safety Report | Annually |
| Other Aggregate Analyses | At time of ISS sponsor submission to any body |
| (any report containing safety data generated during | governing research conduct (e.g., RA, IRB, etc.) |
| the course of the study) | |
| Final (End of Study) Report, including: | At time of ISS sponsor submission to any body |
| <ul> <li>Unblinding data for blinded studies</li> </ul> | governing research conduct (e.g., RA, IRB, etc.) |
| <ul> <li>Reports of unauthorized use of a</li> </ul> | but no later than 1 calendar year after study |
| marketed product | completion |

Aggregate reports should be submitted via email to the Amgen NASCRT manager, accompanied by the Fax Cover Form.

Please refer to the ICH Guidelines E2A for safety related definitions and terminology: http://www.ich.org/fileadmin/Public\_Web\_Site/ICH\_Products/Guidelines/Efficacy/E2A/Step4/E2A\_Guideline.pdf.

#### Accidental Exposures to Talimogene Laherparepvec and Herpetic Event Reporting

In order to better assess and understand the potential risks to treated patients and/or third parties following the treatment of clinical trial subjects with talimogene laherparepvec, special reporting procedures apply for accidental exposures to talimogene laherparepvec and for suspected herpetic events. See Table 4 'Accidental Exposure and Herpetic Event Reporting Requirement Summary.' Clinicians should review the Imlygic package insert (available online) for additional information on the safe handling of talimogene laherparepvec.

# Accidental Exposure of HCPs to Talimogene Laherparepvec

HCPs involved in your clinical trial who were directly exposed to talimogene laherparepvec (e.g., needle stick, splash back) but who are without signs or symptoms of herpetic illness should be reported to Amgen at 1-855-IMLYGIC (1-855-465-9442).

# **Suspected Herpetic Events**

# Suspected herpetic events must be reported to Amgen within 24 hours of awareness.

Reporting is required for: (1) suspected herpetic events in treated patients; (2) suspected herpetic events in at risk HCPs with direct or indirect exposure and 3) suspected herpetic events in treated patient's close contacts, as outlined in Table 4.

In addition to reporting these events, suspected herpetic lesions should be swabbed and submitted for qPCR testing for the detection of talimogene laherparepvec. Samples should be collected using appropriate technique and a flocked swab from site supplies. This test is likely to be more reliable if performed within the **first three days of symptom appearance**. Amgen does not require qPCR or other testing for wild type HSV-1.

#### o Reporting Process for ISS Treated Patients:

- Any suspected herpetic lesion should be reported to Amgen at 1-855-IMLYGIC (1-855-465-9442), evaluated by the Sponsor/Investigator and swabbed for qPCR testing.
- Once an initial report has been made, additional materials will be provided, including reporting forms and supplies needed for shipment of swab samples. Amgen will require patient consent for qPCR testing, which must be obtained prior to swabbing.

#### o Reporting Process for HCPs and Close Contacts:

- Sponsor Investigator should advise any HCPs and/or Close Contacts with suspected herpetic lesions to contact their personal physician to facilitate reporting to Amgen. Suspected herpetic lesions should be reported by the personal physician or exposed individual to Amgen at 1-855-IMLYGIC (1-855-465-9442). Once an initial report has been made, additional materials will be provided, including reporting forms and

supplies needed for the shipment of swab samples. Amgen will require patient consent for qPCR testing, which must be obtained prior to swabbing.

Table 4. Accidental Exposure and Herpetic Event Reporting Requirement Summary

| Exposed<br>Person | Reporter | Timeframe<br>for Reporting<br>to Amgen | Report<br>Mechanism | Timing of<br>Swab<br>Collection | qPCR Testing<br>Required? | Responsible<br>Party for<br>Lesion<br>Swabbing | qPCR Test<br>Result<br>Distribution* |
|---|---|---|---|---|---|---|---|
| Treated Patients with suspected herpetic lesions | Sponsor /<br>Investigator | Within 24<br>hours of<br>Sponsor /<br>Investigator<br>awareness | Contact<br>Amgen at 1-<br>855-IMLYGIC<br>(1-855-465-<br>9442) to report<br>event | Collect swabs<br>from<br>suspected<br>lesions (ideally<br>within 3 days<br>of appearance<br>of symptoms) | Yes, if consent obtained | Sponsor /<br>Investigator | Sponsor /<br>Investigator<br>and Amgen |
| HCP directly<br>exposed to<br>product (e.g.,<br>needle stick,<br>splash back)<br>without signs<br>or symptoms<br>of herpetic<br>illness | HCP's Personal Physician or impacted person | Within 24<br>hours of<br>Reporter<br>awareness | Contact<br>Amgen at 1-<br>855-IMLYGIC<br>(1-855-465-<br>9442) to report<br>event | N/A | N/A | N/A | N/A |
| HCP directly or indirectly exposed to product with suspected herpetic lesions | HCP's<br>Personal<br>Physician or<br>impacted<br>person | Within 24<br>hours of<br>Reporter<br>awareness | Contact<br>Amgen at 1-<br>855-IMLYGIC<br>(1-855-465-<br>9442) to report<br>event | Collect swabs<br>from<br>suspected<br>lesions (ideally<br>within 3 days<br>of appearance<br>of symptoms) | Yes, if consent obtained | HCP or HCP's<br>Personal<br>Physician | HCP's<br>Personal<br>Physician and<br>Amgen |
| Close Contact (eg caregiver, spouse, child) with suspected herpetic lesions | Close<br>Contact's<br>Personal<br>Physician or<br>Close Contact | Within 24<br>hours of<br>Reporter<br>awareness | Contact Amgen at 1- 855-IMLYGIC (1-855-465- 9442) to report event | Collect swabs<br>from<br>suspected<br>lesions (ideally<br>within 3 days<br>of appearance<br>of symptoms) | Yes, if consent<br>obtained | Close<br>Contact's<br>Personal<br>Physician | Close<br>Contact's<br>Personal<br>Physician and<br>Amgen |

# Reporting to the FDA

It is the responsibility of the IND sponsor-investigator to comply with IND safety reporting as set forth in the Code of Federal Regulations, Section 312.32. This responsibility includes providing an annual IND report to the FDA. In addition:


• The FDA will be notified via phone (800-332-1088) or fax (800-FDA-0178) within 7 calendar days of any SAE that is associated with study treatment, is unexpected, andis fatal or life- threatening.

• The FDA will be notified via fax (800-FDA-0178) or online submission (<a href="http://www.fda.gov/downloads/AboutFDA/ReportsManualsForms/Forms/UCM048334.pdf">http://www.fda.gov/downloads/AboutFDA/ReportsManualsForms/Forms/UCM048334.pdf</a>) with a MedWatch (3500A or 3500) within 15 calendar days of any SAE that is associated with the study treatment, unexpected, and serious but not fatal or life-threatening. This includes any previous SAEs that were not initially deemed reportable, but are later determined to meet the criteria for reporting (i.e. by the DSMC).

MedWatch 3500a Reporting Guidelines:

http://www.fda.gov/Safety/MedWatch/HowToReport/DownloadForms/ucm2007307.htm

In addition to completing appropriate patient demographic and suspect medication information, the report should include the following information within the Event Description (section 5) of the MedWatch 3500a form:

- Treatment regimen (dosing frequency, combination therapy)
- Protocol description (and number, if assigned)
- Description of event, severity, treatment, and outcome, if known
- Supportive laboratory results and diagnostics
- Investigator's assessment of the relationship of the adverse event to each investigational product and suspect medication

#### 8. PHARMACEUTICAL INFORMATION

## 8.1 Study Drug: Talimogene Laherparepvec

Talimogene laherparepvec is an oncolytic immunotherapy based on herpes simplex virus type 1 (HSV-1) which is capable of generating an immune response specific to a subject's tumor. Talimogene laherparepvec induces viral lysis of tumor cells, followed by stimulation of a tumor-specific immune response. The following dosage strengths will be made available:

- Talimogene laherparepvec at nominal concentration of 10<sup>6</sup> plaque forming units (PFU)/mL with approximately 1.15 mL in a 2 cc vial for the initial dose
- Talimogene laherparepvec at nominal concentration of 10<sup>8</sup> PFU/mL with approximately 1.15 mL in a 2 cc vial for the second and subsequent doses

#### 8.1.1 Packaging and Formulation of Investigational Product

Talimogene laherparepvec will be presented as a sterile, semi-translucent to opaque solution for injection (opacity is different for each concentration) preservative-free frozen liquid in a single use 2 mL cyclic olefin polymer (COP) plastic resin vial. Each vial will contain talimogene laherparepvec at a nominal concentration of 10<sub>6</sub> PFU/mL or 10<sub>8</sub> PFU/mL in an aqueous sodium phosphate buffer with sodium


chloride, sorbitol and myo-inositol added as stabilizers and water for injection (WFI). Vials are appropriately filled to ensure that a sufficient deliverable dose is provided. Each 2 mL vial will contain approximately 1.15 mL of talimogene laherparepvec with a 1.0 mL deliverable volume. Each vial is intended for single use only and will be available in one of two different presentations:

Current supplies of talimogene laherparepvec is provided as a preservative-free solution in a single—use vial without a clear copolyester plastic sleeve. The product label is found on the vial itself



Future supplies of talimogene laherparepvec will be provided as a preservative-free solution in a single—use vial permanently inserted into a clear copolyester plastic sleeve. The product label will be found on the vial sleeve



Note that the Closed System Transfer Device (CSTD) tested for use with the vial sleeve is the PhaSeal CSTD

Vials will be sealed with gray rubber stoppers, Fluoropolymer-coated on the product side. The vial caps will be color coded and may be used to help distinguish between the 10<sub>6</sub> PFU/mL and 10<sub>8</sub> PFU/mL vial concentrations. The supply for 10<sub>6</sub> PFU/mL vials will be packaged separately from the supply for the 10<sub>8</sub> PFU/mL vials.

- ☐ The 106 PFU/mL strength is supplied in a box containing 10 vials.
- □ The 10<sub>8</sub> PFU/mL strength is supplied in a box containing 20 vials.

The dimensions of the box (of both strengths) are approximately 12.7 x 12.7 x 5 cm (4.891 in. x 4.891 in. x 1.969 inches). Due to the temperature at which talimogene laherparepvec packaging occurs no tamper-evident seal or closure seal will appear on the boxes. Talimogene laherparepvec is sensitive to light and should be protected from light during storage.

#### 8.1.2 Drug storage

To ensure stability and quality are maintained, the product must be stored correctly upon receipt and for the duration of the study under the conditions specified below.

Talimogene laherparepvec must be stored in a non-cycling freezer maintained at a set point of -80°C in a secured location until planned use. Cycling, frost-free, auto defrost freezers must not be used since they cycle to warmer temperatures several times a day. Vials should be kept within the secondary container to protect from light. <u>Table 3</u> outlines the storage temperature requirements.

Storage of Talimogene Laherparepvec - Freezer Set Point

| Freezer Set Point (°C) | Acceptable<br>Variation | Acceptable<br>Range |
|------------------------|-------------------------|---------------------|
| -80°C | ± 10°C | -90°C to -70°C |

Talimogene laherparepvec is stable if maintained in accordance with the guidelines described in this document and the provided expiration date.

To ensure GCP compliance with regards to the storage of biological products, talimogene laherparepvec should be segregated and stored on its own shelf in the

freezer. Sites should also refer to local guidance on storing clinical trial drugs.

#### 8.1.3 Agent Ordering and Agent Accountability

Sponsors of clinical studies are required to establish a record of receipt, storage, use and disposition of all talimogene laherparepvec used to conduct a clinical study. The Sponsor of the clinical study is responsible for ensuring that accountability is maintained and accurate at each clinical site where the study is conducted. At study activation or as required, initial shipments of talimogene laherparepvec 10<sup>6</sup> PFU/mL and 10<sup>8</sup> PFU/mL concentrations will be shipped to the contact and address provided by the Study Sponsor. It is the responsibility of the Study Sponsor to maintain the records of talimogene laherparepvec accountability in accordance with ICH GCP.

Complete study drug information (including packaging, labeling, ordering, storage and disposition) is provided in the Talimogene laherparepvec Pharmacy Information Guide.

#### 9. CORRELATIVE, AND SPECIAL STUDIES

The underlying hypothesis driving this clinical trial is that the induction of high titers of antibody by intra-tumoral talimogene laherparepvec will result in enhanced tumor recognition by the immune system, and subsequently leading to improved disease control. Patients treated on this study will undergo evaluation of immune response to treatment, including serologic response, and evaluation of the baseline and post-treatment cytokine profile and inflammatory response.


The results will be used to correlate response to vaccination with subsequent clinical outcome.

## **Blood Samples:**

Patient serologic and inflammatory response will be measured at baseline during Screening or prior to the Visit Week 1 injection of the study drug, and immediately preceding injections at Visit Weeks 4, 8, 12 or 13

With each collection, 1 Red top tube and 1 pink top tube for serum and mononuclear cells (MNC) will be collected for the following tests:

- Cytokine Profile: IL-1*β*, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12, TNF-alpha, IFN-gamma, IFN-alpha, GM-CSF.
- NK-cell functional assay.

## **Tumor Tissue Samples:**

The tumor biopsy samples will be used to study the relationship between the immune response induced by talimogene laherparepvec and clinical response or resistance to talimogene laherparepvec. Tumor slides will be systemically analyzed at baseline and post-treatment to evaluate changes in the number and/or type of immune cells infiltrating the tumor during treatment. The protocol may be modified to include analysis of the immune and cancer cells in the tumor to identify ribonucleic acid transcripts and/or proteins whose levels change with treatment, and to assess tumor specific mutations or epigenetic changes.

- The biopsy sample will be assessed for baseline tumor infiltrating lymphocytes (TILs) by the same pathologist. This will include CD3, CD4, CD8, CD56, and FOXP3 positive cells.
- Post treatment TILs, as above, will be assessed on the resected tumor at the end of treatment.
- Optional pre- treatment tumor biopsies will be taken from approximately 5 subjects total and immune markers will be compared between pre and post treatment tissue in the immunology lab

Additionally, blood samples and tumor samples may be saved for any potential additional or future analyses such as tumor specific mutations or epigenetic changes (eg, somatic mutations) on tumor tissues.

The study may be amended to include additional testing to ensure analytical methods produce reliable and valid data throughout the course of the study. This can also include, but is not limited to, investigation of unexpected results, incurred sample reanalysis, and analyses for method transfer and comparability.

# 10. STUDY CALENDAR

# 10.1 Study Procedures

| | | | | | | S | tudy | Treati | nent | (week | number | r) <sup>a</sup> | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study<br>Procedures | Screen-<br>ing | 1 <sup>i</sup> | 2 | 3 | 4 <sup>i</sup> | 5 | 6 | 7 <sup>i</sup> | 8 | 9 | 10 <sup>i</sup> | 11 | 12<br>(End of<br>treatment<br>i | Surgery<br>(wks 12-<br>14) | Safety<br>follow<br>up (30<br>days post<br>last<br>TVEC) | Long-<br>term<br>follow<br>up <sup>h</sup> |
| | | | 1 | | | | , | Gener | al Ass | sessm | ents | | T | | | |
| <b>Progress Note</b> | X | X | | | X | X | X | X | X | X | X | X | X | | X | |
| Optional<br>tumor biopsy <sup>k</sup> | X | | | | | | | | | | | | | | | |
| Recording of<br>Concomitant<br>Medications | X | X | | | X | X | X | X | X | X | X | X | X | | X | |
| Vital Signs <sup>b</sup> | X | X | | | X | X | X | X | X | X | X | X | X | | X | |
| Physical<br>Exam,<br>including<br>weight | X | X | | | X | X | X | X | X | X | X | X | X | | X | |
| ECG | X | | | | | | | | | | | | | | | |
| ECOG<br>Performance<br>Status | X | | | | | | | | | | | | | | | |
| Review of AEs<br>& SAEs c | | X | | | X | X | Х | X | Х | X | X | X | X | | X | |
| Talimogene<br>laherparepvec<br>injection <sup>j</sup> | | X | | | X | X | X | X | X | X | X | X | X | | | |
| Correlative<br>labs <sup>i</sup> | | X | | | X | | | | X | | | | X | | | |
| Radiation | | | | | X | X | X | X | X | | | | | | | |
| Survival<br>Status/Disease<br>Recurrence | | | | | | | | | | | | | | | | X |
| | | | | | | | Lo | cal La | bora | tory 1 | Tests d | | | | | |
| Pregnancy<br>(serum or<br>urine) | X | | | | | | | | | | | | | | X | |
| CMP d | X | X | | | X | X | X | X | X | X | X | X | X | | X | |
| CBC,<br>differential,<br>Platelets <sup>d</sup> | X | X | | | X | X | X | Х | X | X | X | Х | X | | X | |
| Coagulation<br>(PT or INR<br>and PTT or<br>aPTT) | X | | | | | | | | | | | | | | | |
| AST, ALT,<br>AlkPhos, Bili,<br>Albumin <sup>d</sup> | X | X | | | X | X | X | X | X | X | X | X | X | | X | |
| TSH, free T3,<br>T4 | X | | | | | | | | ]<br> | | | | | | | |
| | | | | ( | Clinica | 1 & R | adiog | graphi | c Tur | nor/R | esponse | Asses | sments | | | |
| Tumor biopsy | | | | | Mus | t be b | iopsy | confi | rmed | withi | n 3 mon | ths pri | or to stud | y enrollmen | it | |
| Primary<br>Tumor<br>Assessment<br>(MRI/CT) <sup>e, g</sup> | X | | | | | | | | | | | | X | | | |
| CT Chest,<br>Abdomen, | X | | | | | | | | | | | | X | | | |

| Pelvis f |
|----------|

- a. Assessments will occur on Day 1 (+/- 3 days) of the week number.
- b. Blood pressure, resting pulse, respiration rate, and temperature.
- c. All serious adverse events (SAEs) will be reported within 24 hours of the discovery of the event.
- d. May be monitored more frequently if indicated.
- e. Tumor assessment will be documented per RECIST.
- f. CT chest, abdomen, and pelvis at screening (up to 28 days prior to initiation of treatment) and Week 12 (End of treatment)
- g. Primary tumor (MRI/CT) at screening (up to 28 days prior to initiation of treatment) ) and on Day 1 week 12 (± 2 weeks). Simulation scans done for radiation planning are acceptable
- h. Follow up per standard of care (approximately every 12-16 weeks), at the discretion of the treating physician and as per NCCN guidelines. Data for survival status and disease recurrence only will be collected through chart review.
- i. Correlative labs for serologic and inflammatory response; 1 Marble Red top and 1 Pink top. See Section 9 (+/- 7 days).
- j. Talimogene laherparepvec will be given weeks 1 through 12 (+/- 2 weeks) when surgery is expected to be performed. The injections must be given the same day of the week +/- 3 days.
- k. Optional tumor biopsy can be done anytime before week 1 dosing

# **10.2** Screening Procedures:

- Procedures to be completed within 28 days of enrollment/randomization and prior to first treatment (unless otherwise noted).
  - Informed Consent
  - o Review of eligibility criteria
  - o Recording of medical history and concomitant medications
  - Physical Exam (including weight)
  - o ECG
  - Vital Signs (Blood pressure, resting pulse, respiratory rate, temp.)
  - o Radiographic imaging (Chest, abdomen, and pelvis and all other sites of disease)
  - o Imaging of primary tumor site
- Laboratory Assessments
  - o Within 28 days of enrollment and prior to first treatment.
    - HIV test: Required if clinically indicated
    - Hepatitis B and/or C tests: Required if clinically indicated
  - $\circ$   $\leq 10$  days of enrollment
    - Hematology panel (with 5 part differential). 3 part differential if 5 part unable to be performed.
    - Chemistry panel
    - Coagulation panel
    - Thyroid function tests
  - $\circ \le 3$  days of enrollment
    - Serum or urine pregnancy test for females of childbearing potential

## 10.3 Long-term Follow up

After the end of treatment visit is completed, subjects will be followed according to standard of care (approximately every 12 weeks), at the discretion of the treating physician, at which time disease recurrence and survival status will be assessed for up to 5 years. Data for disease recurrence and survival status only will be collected per chart review, phone call or email.

#### 11. MEASUREMENT OF EFFECT

## 11.1 Pathologic Response

At the end of the neoadjuvant therapy, patients will undergo resection of the treated tumor. The pretreatment biopsy and all the resected tumor samples must be reviewed by the same pathologist.

- The percentage of post treatment tumor necrosis must be documented. The primary end point for this study is pathologic complete response (pCR) and is defined as ≥ 90% tumor necrosis following concurrent radiation therapy and talimogene laherparepyec.
- Additional immunohistochemical studies will be performed as described in Section 9.

## 11.2 Time to Disease progression (TTP)

TTP is defined as the time from Enrollment until objective tumor progression including local and distant recurrences.

## 11.3 Other Response Parameters

The following response assessment guidelines may be amended during the course of the study if changes are made to the current RECIST Guidelines or if a new disease assessment tool becomes available.

#### Response Measurement Criteria:

- Measurements of the tumor in its largest dimension should be obtained at baseline and at the end of the treatment phase, prior to surgical resection.
- Response criteria should be by RECIST.
  - Complete response is the disappearance of all target lesions.
  - Partial response is a 30% decrease in the sum of the longest dimensions of the target lesions, relative to baseline.
  - Progressive disease is an increase of 20% or more in the sum of the longest dimension of target lesions
  - Stable disease is a decrease in the tumor size of < 30% or an increase of < 20%.
- Antitumor response by pathologic assessment will be performed on the resected tumors.
- Pathologic assessment will be performed per institutional guidelines.
  - The percent of tumor necrosis and the percent of tumor-infiltrating lymphocytes will be documented.
  - Complete pathological response will be considered ≥ 90% pathologic tumor necrosis.

Radiologic response will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) [Eur J Ca 45:228-247, 2009]. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the


RECIST criteria.

Please see Appendix B for more details of the RECIST Guidelines.

#### 12. STATISTICAL CONSIDERATIONS

#### 12.1 Study Design/Endpoints

#### Phase Ib

| Thase ID | |
|---|---|
| The primary objectives of this Phase Ib | Decision Rule |
| study are to 1) assess safety and | |
| tolerability, and to 2) determine the | |
| recommended Phase II dose of | |
| neoadjuvant administration of | |
| talimogene laherparepvec in | |
| combination with external beam | |
| radiation therapy in the treatment of | |
| soft tissue sarcoma. An initial cohort of | |
| 3 patients will be treated at dose level | |
| 0. Decisions on when and how to dose | |
| de-escalate are described below. | |
| Number of Patients with DLT at a | |
| Given Talimogene Laherparepvec | |
| Dose | |
| $\geq 2$ | Dose level will be declared toxic. |
| | If this is the lowest dose level, stop the study due to |
| | excessive toxicity; otherwise enter <i>three</i> additional |
| | patients at the next lowest dose level. |
| $\leq 1$ out of 3 | Enter <i>three</i> more patients at this dose level. |
| $\leq 1$ out of 6 | This is the recommended Phase II dose. |

Up to 6 patients will be treated at each dose level. The recommended Phase II dose will be defined as the highest dose level for which at most 1 out of 6 patients experience a DLT.

#### Phase II

The primary objective of the Phase II portion of this study is to evaluate the preliminary evidence of anti-tumor activity of talimogene laherparepvec in combination with external beam radiation therapy. The primary endpoint of interest is pathologic complete response (pCR) rate defined as the proportion of subjects with pathologic tumor necrosis of  $\geq 90$  %. Estimates of historic pCR based on tumor necrosis  $\geq 90$ % for the treatment of soft tissue sarcomas with external beam radiation therapy are not available in the current literature. However, a pCR rate of 30% would be considered unacceptable for the proposed combination treatment whereas a pCR of 55% or more is considered clinically important. Sample size requirements are based on an optimal Simon two-stage design with 80% power and a significance level of 5%. Nine (9) patients will

be enrolled in the first stage, and the study will be terminated if 3 or fewer respond. Otherwise, an additional 26 patients will be enrolled in the second stage. If 15 or more of the 34 total patients respond, the treatment will be deemed worthy of further investigation. This design has an expected sample size of 16.0 and a 0.73 probability of early termination.

## **Data Analysis and Reporting**

The number and severity of all adverse events will be summarized by simple descriptive statistics. pCR and ORR (CR+PR) rate point estimates and 95% exact confidence intervals will be reported. For TTP (time from first day of study treatment to first documented disease progression) and OS (time from first day of study treatment to death due to any cause), survival curves using the Kaplan-Meier method will be constructed. Estimates along with 95% confidence intervals will be reported.

#### **REFERENCES**

- 1. Siegel R, Naishadham D, Jemal A. Cancer Statistics 2012. CA Cancer J Clin. 2012 Jan-Feb;62(1):10-29. doi: 10.3322/caac.20138. Epub 2012 Jan 4
- 2. National Comprehensive Cancer Network (NCCN). Clinical Practice Guidelines In Oncology: Soft Tissue Sarcoma Vol2. 2012. www.nccn.org.
- 3. Pisters PWT, Leung DHY, Woodruff J, Shi W, and Brennan MF. Analysis of Prognostic Factors in 1,041 Patients With Localized Soft Tissue Sarcomas of the Extremities. J Clin Oncol, Vol 14, No 5 (May), 1996: pp 1679-1689
- 4. Rosenberg S, Tepper J, Glatstein E, et al: The treatment of soft-tissue sarcomas of the extremities: Prospective randomized evaluations of (1) limb-sparing surgery plus radiation therapy compared with amputation and (2) the role of adjuvant chemotherapy. Ann Surg 196:305-315, 1982
- 5. Yang J, Chang A, Baker A, et al: Randomized prospective study of the benefit of adjuvant radiation therapy in the treatment of soft tissue sarcomas of the extremity. J Clin Oncol 16:197-203, 1998
- 6. Pisters P, Harrison L, Leung D, et al: Long-term results of a prospective randomized trial of adjuvant brachytherapy in soft tissue sarcoma. J Clin Oncol 14:859-868, 1996
- 7. Canter RJ, Martinez SR, Tamurian RM, et al. Radiographic and histologic responseto neoadjuvant radiotherapy in patients with soft tissue sarcoma. Ann Surg Oncol. 2010 Oct;17(10):2578-84
- 8. Shah D, Borys D, Martinez SR, et al. Complete pathologic response to neoadjuvant radiotherapy is predictive of oncological outcome in patients with soft tissue sarcoma. Anticancer Res. 2012 Sep;32(9):3911-5.
- 9. O'Sullivan B, Davis A, Turcotte R, et al: Preoperative versus postoperative radiotherapy in soft-tissue sarcoma of the limbs: A randomized trial. Lancet 359:2235-2241, 2002
- 10. Davis A, O'Sullivan B, Turcotte R, et al: Late radiation morbidity following randomization to preoperative versus postoperative radiotherapy in extremity soft tissue sarcoma. Radiother Oncol 75:48-53, 2005

- 11. Cannon CP, Ballo MT, Zagars GK, et al. Complications of combined modality treatment of primary lower extremity soft-tissue sarcomas. Cancer 2006;107:2455–2461.
- 12. Cheng EY, Dusenbery KE, Winters MR, et al. Soft tissue sarcomas: Preoperative versus postoperative radiotherapy. J Surg Oncol 1996;61:90–99.
- 13. San Miguel I, San Julian M, Cambiero M, et al. Determinants of toxicity, patterns of failure, and outcome among adult patients with soft tissue sarcomas of the extremity and superficial trunk treated with greater than conventional doses of perioperative high-dose rate Brachytherapy and external beam radiotherapy. Int. J. Radiation Oncology Biol. Phys., Vol. 81, No. 4, pp. e529–e539, 2011
- 14. Devisetty K, Kobayashi W, Suit HD, et al. Low-dose neoadjuvant external beam radiation therapy for soft tissue sarcoma. Int. J. Radiation Oncology Biol. Phys., Vol. 80, No. 3, pp. 779–786, 2011
- 15. Lee S, Obata Y, Yoshida M, et al. Immunomic analysis of human sarcoma. Proc Natl Acad Sci U S A. 2003 Mar 4;100(5):2651-6. Epub 2003 Feb 24.
- 16. Segal NH, Blachere NE, Shiu HYA, et al. Antigens recognized by autologous antibodies of patients with soft tissue sarcoma. Cancer Immunity, 2005; 5:1424-9634
- 17. Jungbluth A, Antonescu C, Busam K, et al. Monophasic and biphasic synovial sarcomas abundantly express cancer/testis antigen NY-ESO-1 but not MAGE-A1 or CT7. Int J Cancer. 2001 Oct 15;94(2):252-6.
- 18. Newman W, Southam C. Virus treatment in advanced cancer; a pathological study of fifty-seven cases. Cancer 1954;7:106-18.
- 19. Papanastassiou V, Rampling R, Fraser M, et al. The potential for efficacy of the modified (ICP 34.5(-)) herpes simplex virus HSV1716 following intratumoural injection into human malignant glioma: a proof of principle study. Gene Ther 2002;9:398-406.
- 20. Rampling R, Cruickshank G, Papanastassiou V, et al. Toxicity evaluation of replication-competent herpes simplex virus (ICP 34.5 null mutant 1716) in patients with recurrent malignant glioma. Gene Ther 2000;7:859-66.
- 21. Kanai R, Tomita H, Hirose Y, et al. Augmented therapeutic efficacy of an oncolytic herpes simplex virus type 1 mutant expressing ICP34.5 under the transcriptional control of musashi1 promoter in the treatment of malignant glioma. Hum Gene Ther 2007;18:63-73.
- 22. Kohno SI, Luo C, Nawa A, et al. Oncolytic virotherapy with an HSV amplicon vector expressing granulocyte-macrophage colony-stimulating factor using the replication-competent HSV type 1 mutant HF10 as a helper virus. Cancer Gene Ther 2007;14:918-26.
- 23. Finkelstein SE, Iclozan C, Bui MM, et al. Combination of external beam radiotherapy (EBRT) with intratumoral injection of dendritic cells as neo-adjuvant treatment of high-risk soft tissue sarcoma patients. Int J Radiat Oncol Biol Phys. 2012 Feb 1;82(2):924-32.
- 24. Hiniker SM, Chen DS, Knox SJ. Abscopal effect in a patient with melanoma. N EnglJ Med. 2012 May 24;366(21):2035
- 25. Postow MA, Callahan MK, Barker CA. Immunologic correlates of the abscopal effect in a patient with melanoma. N Engl J Med. 2012 Mar 8;366(10):925-31.
- 26. Harrington K, Hingorani M, Tanay MA, et al. Phase I/II study of oncolytic HSVGM-CSF in combination with radiotherapy and cisplatin in untreated stage III/IV squamous cell cancer of the head and neck. *Clin Cancer Res.* 2010;16:4005-4015.


- 27. Hu J, Coffin R, Davis C. A phase I study of oncovexGM-CSF, a second-generation oncolytic herpes simplex virus expressing granulocyte macrophage colony-stimulating factor. Clin Cancer Res 2006;12:6737-6747.
- 28. ClinicalTrials.gov.
- 29. Senzer NN, Kaufman HL, Amatruda T, et al. Phase II clinical trial of a granulocytemacrophage colony-stimulating factor-encoding, second-generation oncolytic herpesvirus in patients with unresectable metastatic melanoma. J Clin Oncol. 2009;27(34):5763-5771.
- 30. Small, EJ, Schellhamer, PF, Higano, C, et al. Immunotherapy (APC8015) for androgen independent prostate cancer (AIPC): final survival data from a phase 3 randomized placebo-controlled study. Amer Soc Clin Oncol,: abstract #264, 2005

# APPENDIX A PERFORMANCE STATUS CRITERIA

| ECC | OG Performance Status Scale | Karnofsky Performance Scale | |
|---|---|---|---|
| Grade | Descriptions | Percent | Description |
| 0 | Normal activity. Fully active, able to carry on all pre-disease | 100 | Normal, no complaints, no evidence of disease. |
| | performance without restriction. | 90 | Able to carry on normal activity; minor signs or symptoms of disease. |
| 1 | Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able | 80 | Normal activity with effort; some signs or symptoms of disease. |
| 1 | to carry out work of a light or sedentary nature ( <i>e.g.</i> , light housework, office work). | Cares for self, unable to carry on normal activity or to do active wor | |
| 2 | In bed <50% of the time. Ambulatory and capable of all self-care, but unable to carry out | 60 | Requires occasional assistance, but is able to care for most of his/her needs. |
| | any work activities. Up and about more than 50% of waking hours. | 50 | Requires considerable assistance and frequent medical care. |
| 3 | In bed >50% of the time. Capable of only limited self-care, confined | 40 | Disabled, requires special care and assistance. |
| 3 | to bed or chair more than 50% of waking hours. | 30 | Severely disabled, hospitalization indicated. Death not imminent. |
| 4 | 100% bedridden. Completely disabled. Cannot carry on any | 20 | Very sick, hospitalization indicated. Death not imminent. |
| 4 | self-care. Totally confined to bed or chair. | 10 | Moribund, fatal processes progressing rapidly. |
| 5 | Dead. | 0 | Dead. |


APPENDIX B RECIST GUIDELINES

 $\underline{http://www.eortc.be/recist/documents/RECISTGuidelines.pdf}$ 


**APPENDIX C:** CTCAE V.4.0

http://evs.nci.nih.gov/ftp1/CTCAE/CTCAE\_4.03\_2010-06-14\_QuickReference\_5x7.pdf

#### APPENDIX D: CONTRAINDICATIONS AND ADVERSE EVENTS

#### CONTRAINDICATIONS

Talimogene laherparepvec is contraindicated in patients with a history of life-threatening hypersensitivity to talimogene laherparepvec or any of its excipients.

## **ADVERSE DRUG REACTIONS**

#### **Gastrointestinal disorders SOC:**

Very Common ( $\geq 10\%$ )

• Nausea, Vomiting, Diarrhea, Constipation

Common ( $\geq$ 1% and  $\leq$ 10%)

• Weight loss

#### General disorders and administrative site condition SOC:

Very Common (≥ 10%)

• Chills, Pyrexia, Fatigue, Flu like symptoms, Injection site pain

Common ( $\geq$ 1% and  $\leq$ 10%)

• Injection site reactions (including erythema, inflammation, warmth, pain [at injection site and at distant, non-injected lesions], swelling [at injection site and/or lymphadenopathy], or drainage may occur), Malaise

#### Metabolism and nutrition disorders SOC:

Common ( $\geq$ 1% and  $\leq$ 10%)

Dehydration

#### Blood and lymphatic system disorders SOC:

Common ( $\geq$ 1% and  $\leq$ 10%)

• Anemia

Uncommon ( $\geq 0.1\%$  and < 1%)

• Plasmacytoma at the injection site

#### Musculoskeletal and Connective tissue disorders SOC:

Very Common (≥ 10%)

• Myalgia, Arthralgia, Pain in extremity

#### **Infections and Infestations SOC:**

Common ( $\geq$ 1% and  $\leq$ 10%)

• Cellulitis (see Warnings and Precautions), Oral herpes

Uncommon ( $\geq 0.1\%$  and < 1%)

• Delayed wound healing


## Injury, poisoning and procedural complications:

Common ( $\geq$ 1% and  $\leq$ 10%)

• Bruising

#### **Vascular disorders SOC:**

Common (≥1% and <10%)

• Flushing

## **Nervous System Disorder SOC:**

Very Common (≥ 10%)

Headache

Common ( $\geq$ 1% and  $\leq$ 10%)

Dizziness

#### Skin and subcutaneous tissue disorders SOC:

Common ( $\geq$ 1% and  $\leq$ 10%)

• Vitiligo

## Respiratory, thoracic and mediastinal disorders SOC:

Uncommon ( $\geq 0.1\%$  and < 1%)

• Laryngeal swelling

#### EFFECTS ON ABILITY TO DRIVE AND USE MACHINES

None known.

#### **OVERDOSE**

The maximum dose of talimogene laherparepvec that can be safely administered has not been determined.

#### ABUSE AND DEPENDENCE

Talimogene laherparepvec is not a controlled substance. There is no evidence that talimogene laherparepvec is habit forming or could lead to dependence.

#### PEDIATRIC USE

No studies of talimogene laherparepvec have been conducted in pediatric subjects.

#### **GERIATRIC USE**

There are subjects > 65 as well as > 75 years of age who have received talimogene laherparepvec. However, no adequate and well-controlled studies have been designed to specifically evaluate the use of talimogene laherparepvec in geriatric subjects.

#### RENAL IMPAIRMENT

No clinical studies have been conducted in patients with severe renal impairment.

#### **HEPATIC IMPAIRMENT**


No clinical studies have been conducted in patients with severe hepatic impairment.


# APPENDIX E: DATA AND SAFETY MONITORING PLAN Type of Clinical Trial:

**X** Investigator-initiated (UI/HCCC) Investigator-initiated, participating site

Pilot study Phase I

X Phase I/II Phase II

Phase III Compassionate-use/Expanded Access

X Interventional Treatment Interventional Non-Treatment

Non-Interventional

## **Study risk-level:**

Level 1—low risk of morbidity or death, \* <1% of death or any adverse event

Level 2—risk of death\* <1% or any adverse event 1% – 5%

Level 3—risk of death\* 1% – 5% or grade 4 – 5 SAE 1% – 5%

X Level 4—risk of death\* >5% or grade 4 – 5 SAE >5% Drugs being used on a "compassionate" basis

## **Reporting and Monitoring Requirements:**

All institutional investigator initiated trials (IITs), regardless of assigned risk level are subject to routine DSMC monitoring activities which may include but are not limited to review of signed consent documents, eligibility and adverse event reporting.

All institutional IITs have the following **reporting requirements** as part of their DSMP:

- Register all subjects in HCCC's Clinical Trial Management System, OnCore
- Document Adverse Events
- Document protocol deviations
- Provide an annual progress report to the DSMC via OnCore data export

## Selected monitoring strategy based on risk-level:

#### Risk Level 4

Interventional treatment trials involving investigational agents or devices with a risk of death\* (>5% or grade 4 – 5 SAE >5%), e.g. all investigator initiated INDs, most Phase I/II

<sup>\*</sup> Risk of death" refers specifically to 100-day treatment-related mortality


trials, gene therapy, gene manipulation or viral vector systems high-risk clinical procedures if performed solely for research purposes. The use of a new chemical or drug for which there is limited or no available safety data in humans.

## Study Safety Review

An independent study monitor and/or the DSMC Chair (or designee), will review study data (provided by the PI/available in OnCore) and communicate with the PI at least biannually. A copy of this communication will be forwarded to the DSMC and PRMC Chairs.

## **Additional Reporting Requirements:**

- A scanned copy of the completed eligibility checklist, with screening information and PI signature, will be attached in OnCore for ongoing review by DSMC staff.
- Serious adverse events will be entered directly into an OnCore SAE report by the research team. OnCore will send an automatic notification to the DSMCChair/acting Chair and staff for review.
- The DSMC utilizes a risk-based monitoring approach. The trial's research records will be monitored at minimum twice per year. Monitoring may be done more frequently depending on the protocol, risks to subjects, reported serious/adverse events, patient population and accrual rate. Records for a minimum of 25% of subjects will be monitored for the entire study.

Monitoring will involve the following:

- review eligibility of patients accrued to the study,
- check for the presence of a signed informed consent,
- determine compliance with protocol's study plan,
- determine whether SAEs are being appropriately reported to internal and external regulatory agencies,
- compare accuracy of data in the research record with the primarysource documents,
- review investigational drug processing and documentation.
- assess cumulative AE/SAE reports for trends and compare to study stopping rules.

# Routine Adverse Event Reporting

For non-serious Adverse Events, documentation must begin from the time the subject signs the informed consent document and continue through the 30-day follow-up period after the last dose of study drug.


Collected information should be recorded in the electronic/Case Report Forms (eCRF/CRF) for that subject. A description of the event, its severity or toxicity grade (according to NCI's Common Toxicity Criteria (CTCAE)), onset and resolved dates (if applicable), and the relationship to the study drug should be included. Documentation should occur in real time. The principal investigator has final responsibility for determining the attribution of the event as it is related to the study drug.

•

## Serious Adverse Event Reporting

For any experience or condition that meets the definition of a serious adverse event (SAE), recording of the event must begin after signing of the informed consent and continue through the 30 day follow-up period after treatment is discontinued.

Investigators must report to the DSMC any serious adverse events (SAE), whether or not they are considered related to the investigational agent(s)/intervention (21 CFR 312.64). SAEs must be reported via an OnCore SAE Report within 24 hours of learning of the event.

An adverse event is considered **serious** if it results in ANY of the following outcomes:

- 1. Death
- 2. A life-threatening adverse event
- 3. An adverse event that results in inpatient hospitalization OR prolongation of existing hospitalization for  $\geq$  24 hours
- 4. A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- 5. A congenital anomaly/birth defect.
- 6. Important Medical Events (IME) that may not result in death, be life threatening, or require hospitalization may be considered serious when, based upon medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. (FDA, 21 CFR 312.32; ICH E2A and ICH E6).

# FDA Reporting Requirements (for Sponsor-Investigators)

It is the responsibility of the IND sponsor-investigator to comply with IND safety reporting as set forth in the Code of Federal Regulations, <u>Section 312.32</u>. This responsibility includes providing an annual IND report to the FDA.

All IND safety reports must be submitted on Form 3500A and be accompanied by Form 1571. The type of report (initial or follow-up) should be checked in the respective boxes on Forms 3500A and 1571. See Instructions for completing Form 3500A. Please note all instance of UIHC, location, and faculty / staff should be redacted from supporting documentation and the 3500A.

#### The submission must be identified as:

- "IND safety report" for 15-day reports, or
- "7-day IND safety report" for unexpected fatal or life-threatening suspected adverse reaction reports, or
- "Follow-up IND safety report" for follow-up information.

For detailed explanation of the above definitions, requirements, and procedures related to IND application safety reports and the responsibilities of IND applications sponsors with regard to such reporting, refer to <u>Guidance for Industry and Investigators</u>: <u>Safety Reporting Requirements for INDs and BA/BE Studies (PDF - 227KB)</u>

In addition to completing appropriate patient demographic and suspect medication information, the report should include the following information within the Event Description (section 5) of the MedWatch 3500A form:

- Treatment regimen (dosing frequency, combination therapy)
- Protocol description (and number, if assigned)
- Description of event, severity, treatment, and outcome, if known (grading the event per CTCAE)
- Supportive laboratory results and diagnostics
- Sponsor-Investigator's assessment of the relationship of the adverse event to each investigational product and suspect medication

## **Data Monitoring and Management**

#### Subject Registration

All studies that undergo PRMC review and/or utilize HCCC Clinical Research Services (CRS) resources are required to register subjects in OnCore. Each subject registration includes the following:

- The subject's IRB approved (version date) consent form and the date of their consent.
- Date of eligibility and eligibility status (eligible, not eligible)
- On study date and subject's disease site (and histology if applicable)
- On treatment date (if applicable)

All subject registration information is expected to be entered into OnCore within **2 (two) business days** after the subject's study visit.


Subject Data

For HCCC investigator initiated trials, research staff are responsible for entering subject study data (data collection) into OnCore electronic case report forms (eCRFs). These eCRFs must be approved by the PI and statistician prior to study activation to ensure sufficient and necessary data acquisition. All information entered into eCRFs will be traceable to the source documents which are generally maintained in the subject's file.

eCRF data entry needs to be timely and should be entered into OnCore as soon as possible but no later than **14 (fourteen) business days** after the subject's visit, including adverse events, tumor measurements, administration of study medication, concomitant medications, labs, and vitals. Physical exam assessments must be entered no later than **14 (fourteen) business days** following completion of the physician's clinic note in the medical record.

Timely data entry facilitates remote monitoring of data, allows the data to progress appropriately through the data cleaning process, and helps prevent a backlog of data queries.

## Forms Monitoring

OnCore eCRF data are monitored on a routine basis (dependent on accrual) to ensure all data are entered completely, accurately, and within time requirements outlined above. The assigned DSMC monitor will coordinate and complete the data monitoring review. When the time comes to monitor a study (based on patient accrual and assigned risk level of trial) the monitor arranges for a selection of cases to be reviewed from among the subjects registered in OnCore. As part of the forms monitoring process, the assigned monitor will issue queries via OnCore (linked to the eCRF) to resolve missing, incomplete, and/or incorrect information. A member of the research team is expected to respond to these monitoring queries within 14 (fourteen) business days.

The monitoring process can often identify misunderstandings or deficiencies in the written, research protocol requirements earlier in the study process and thereby improve data quality and reduce rework.

#### Final Reports

A summary of each subject's data record is continually available to the PI, research staff, and DSMC from OnCore's Biostat Console. The availability of this information is a valuable tool for the preparation of final reports and manuscripts as well as ongoing deficiency reports.

## **Eligibility Checklist**

# Eligibility Checklist

| Si | bject ID: Date: | |
|---|---|---|
| Exclu | sion Criteria. All responses must be marked NO or NA for patient to be eligible | |
| | Certain histologic subtypes: GIST, Desmoid, Ewing sarcoma, Kaposi sarcoma, bone sarcomas and myxoid liposarcomas Grade 1 | Yes No |
| 2. | History or evidence of sarcoma associated with immunodeficiency states (e.g., hereditary immune deficiency, HIV, organ transplant or leukemia) | Yes No |
| 3. | Subject with retroperitoneal and visceral sarcoma | Yes No |
| 4. | History or evidence of gastrointestinal inflammatory boweldisease (ulcerative colitis or Crohn's disease) or other symptomatic autoimmune disease including inflammatory bowel disease or history of any poorly controlled or severe systemic autoimmune disease (e.g., rheumatoid arthritis, systemic lupus erythematosus, scleroderma, type I diabetes, autoimmune vasculitis) | Yes No |
| 5. | History of other malignancy within the past 3 years except iftreated with curative intent and no known active disease present and has not received chemotherapy for $\geq 1$ year before enrollment / randomization and low risk for recurrence. | Yes No |
| 6. | History of prior or current autoimmune disease. | Yes No |
| 7. | History of prior or current splenectomy or splenic irradiation. | Yes No |
| 8. | Active herpetic skin lesions. | Yes No |
| 9. | Require intermittent or chronic treatment with an anti-herpetic drug (e.g., acyclovir), other than intermittent topical use. | Yes No |
| 10 | . Any non-oncology vaccine therapies used for the prevention of infectious disease within 28 days prior to enrollment and during treatment period. | Yes No |
| 11 | . Concomitant treatment with therapeutic anticoagulants such as warfarin. | Yes No |
| 12 | . Known human immunodeficiency virus (HIV) disease (requires a negative test for clinically suspected HIV infection). | Yes No |
| 13 | . Acute or chronic hepatitis B or hepatitis C infection (requires a negative | Yes<br>No |
| | <ul> <li>test for clinically suspected hepatitis B or hepatitis C infection).</li> <li>Evidence of hepatitis B</li> <li>1. Positive HBV surface antigen (indicative for chronic hepatitis B or</li> </ul> | |

2. Negative HBV surface antigen but positive HBV totalcore antibody (indicative for resolved hepatitis B infection or

recent acute hepatitis B)

occult hepatitis B) and detectable copies of HBV DNA by PCR (detectable HBV DNA copies suggest occult hepatitis B).

- Evidence of hepatitis C
  - 1. Positive HCV antibody and positive HCV RNA by PCR (undetectable RNA copies suggest past and resolved hepatitis C infection).

| 14. Female subjects who are pregnant or breast-feeding, or planning to become pregnant during study treatment and through 3 months after the last dose of study treatment. | | Yes No |
|---|---|---|
| 15. Female subjects of childbearing potential or male subjects unwillingto use 2 highly effective methods of contraception during study treatment and through 3 months after the last dose of study treatment. See section 7.5 for more details. | | |
| 16. Currently receiving treatment in another investigational device ordrug study, or less than 30 days since ending treatment on another investigational device or drug study(s). | | |
| 17. Other investigational procedures while participating in this study that co | auld | |
| affect the primary objective of the study as determined by the PI are exc | | Yes No |
| 18. Previously enrolled in this study. | | Yes No |
| 19. Receiving any other investigational agents. | | Yes No |
| 20. Evidence of CNS metastases. | | Yes No |
| 21. History of allergic reactions attributed to compounds of similarchemical biologic composition to talimogene laherparepvec. | l or | Yes No |
| 22. Uncontrolled intercurrent illness including, but not limited to, ongoing of active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness / social situations that would limit compliance with study requirements. | | Yes No |
| 23. Receiving or requiring immunosuppressive therapies. | | Yes No |
| 24. Laboratory abnormalities: | | |
| Hemoglobin < 9.0 g/dL | Yes No | |
| Absolute neutrophil count (ANC) < 1500 per mm <sup>3</sup> | Yes No | |
| Platelet count < 100,000 per mm <sup>3</sup> | Yes No | |
| Total bilirubin > 1.5 X ULN | Yes No | |
| Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) | Yes No | |

 $> 2.5 \times ULN$ 

Alkaline phosphatase > 2.5 x ULN

Creatinine > 2.0 x ULN

PT (or INR) and PTT (or aPTT) > 1.5 x ULN

Yes No

Yes No

Yes No

| Signature: | Date: |
|------------|-------|

# **Expected toxicities**

The following anticipated risks are identified due to this clinical trial:

- Very Common side effects (which may affect more than 1 person in 10):
  - o Flu like illness: chills, fever, feeling tired, muscle pain, nausea and vomiting
  - o Injection site pain
  - Headache
  - Joint pain
  - o Arm or leg pain
  - o Diarrhea
  - Constipation
- Common side effects (which may affect between 1 and 10 people in every 100):
  - Injection site reactions: bleeding, redness, swelling, inflammation
    - Skin infection caused by bacteria at the site of injection; symptoms may include fever, chills, redness or swelling at the injection site or site of the tumor, and may require hospitalization for antibiotic treatment
    - Wound complication at the injection site (secretion or discharge)
    - O Pain: pain after procedure, in the tumor, in the abdomen, throat pain, pain in the armpit or groin
    - Abdominal discomfort
    - Areas of skin with loss of color (Vitiligo)
    - o Cold sore or fever blister in mouth (Oral herpes)
    - o Low red blood cell count (Anemia)
    - Not feeling well (Malaise)
    - Weight loss
    - Dehydration
    - o Bruise
    - Dizziness
    - o Skin or face becomes warm and reddened (Flushing)
- Uncommon side effects (which may affect between 1 and 10 in every 1000):
  - o Injection site reactions: warmth, incision site infection


- O Swelling in the voice box area of your throat that might result in needing a surgical procedure on the neck to open a direct airway. This occurred in a talimogene laherparepvec-treated patient who had a similar problem before treatment. A tube might need to be inserted into the opening in your throat. This tube may be connected to a machine to help you breathe.
- o Plasmacytoma (a collection of abnormal antibody-producing white blood cells) in the area where talimogene laherparepvec is injected. Plasmacytoma may be associated with multiple myeloma (a cancer of plasma cells affecting the bone marrow).
- O Symptoms of delayed wound healing at or around the injection site such as injection site discharge, foul odor, or dead tissue at the injection site. If you notice symptoms of delayed wound healing at the injection site(s), especially if you have risk factors such as diabetes, poor blood circulation, have had radiation to the site, you should contact the study doctor or his/her study staff immediately.

## Other potential side effects

- Allergic Reaction: As with any medication, you may have an allergic reaction to talimogene laherparepvec. Symptoms of an allergic reaction in general may include headache, rash, itching, flushing, swelling, shortness of breath, nausea and sometimes vomiting. Severe allergic reactions can cause dizziness, severe skin reactions, difficulty breathing or swallowing, a decrease in blood pressure, and could be life threatening. If you have symptoms of an allergic reaction, you should contact the study doctor or his/her study staff immediately. If you have had an allergic reaction to talimogene laherparepvec or any of its ingredients, you should inform your doctor.
- Autoimmune Reactions: Autoimmune reactions to the body's own tissues have been reported in some patients administered talimogene laherparepvec. Examples of autoimmune reactions that have been reported in patients receiving talimogene laherparepvec include inflammation of the kidneys (nephritis), blood vessels (vasculitis), lungs (pneumonitis) and worsening psoriasis. It is possible that an autoimmune reaction could occur in any part of the body. Please tell your doctor if you have had any type of autoimmune disease before treatment with talimogene laherparepvec, and all treatments you are receiving for the disease.

# **Stopping Rules:**

As a phase II study, stopping rules do not apply. If a subject dies during active study treatment:

- Trial will be placed on accrual hold until case review
- The death will be reviewed by the principal investigator, IND medical monitor, and IND sponsor (and, as applicable, treating physician)
- Adverse events, including deaths on study, will be reviewed at IND investigators' meeting.

Appendix F

Serious Adverse Drug Reaction

| Investigator Sponsored Study (ISS) FAX Transmittal Form | |
|---|---|
| Talimogene Laherparepvec (T-VEC) | |
| To: Amgen Global Safety Toll-free#:1-888-814-8653 | AMGEN ISS PROTOCOL |
| For countries where the U.S. toll-free | #:20139075 |
| # cannot be used: +44-20-7136-1046 | Sponsor: |
| | 1.1.1.1.1 Sponsor Contact Name: |
| Email ( <u>Only</u> for sponsors with a secure email connection with Amgen): | Fax No: |
| svc-ags-in-us@amgen.com | Phone No: |
| | Date: |
| Use this form as a cover page for an individual listings. | report, for batched individual reports, and for line |
| ***NOTE: Please use data reconciliation fax cov | ver sheet to submit data reconciliation line listings. |
| 1.1.1.1.2 Fax transmission contents (Check all th | at apply): |
| To be sent <u>immediately</u> after each single case submission to RA, EC, IRB or DMC: 1.1.1.1.3 Expeditable Serious Adverse Events/Serious Adverse Drug Reactions # of Reports Submitted: To be sent in regular intervals per contractual agreement (eg, as batched individual reports or line listings): | |
| Serious Adverse Drug Reactions | # of Reports Submitted: |
| Period from to DDMMM/YYYY DD/MMM/YYYY | _ |
| Serious Adverse Events | # of Reports Submitted: |
| (does <u>NOT</u> apply for marketed Amgen products) Period from to DD/MMM/YYYY DD/MMM/YYYY | |
| Other Reports (to be sent as per contractual agreement eg, pregnancy/lactation reports) | |
| Specify type of report: | # of Reports Submitted: |
| Period from to DD/MMM/YYYY | |
| For multi-country studies please indicate c | ountries of transmitted report(s) origin: |

| Total # of pages in this transmission, including cover page: |
|--------------------------------------------------------------|
| , |

Appendix G

Aggregate Safety Reporting
Investigator Sponsored Study (ISS)

FAX Transmittal Form
Imlygic (Talimogene Laherparepvec, T-VEC)

To: NASCR Study Management

Email: dogoldst@amgen.com

AMGEN ISS PROTOCOL #:\_20139075\_\_\_

PI/Sponsor:

1.1.1.3.1 Site Contact Name:

Fax No:\_\_\_\_\_

Phone No:

Date:

Use this form as a cover page for all aggregate safety reporting

| 1.1.1.1.4 Fax transmission contents (Check all that apply): | |
|---|---|
| Description of Reports | |
| 1.1.1.1.5 Adverse Event Line Listing 1.1.1.1.6 (all serious and non-serious events, regardless of relatedness) | |
| 1.1.1.1.7 Adverse Events Summary Tabulation 1.1.1.1.8 (all serious and non-serious events, regardless of relatedness) | |
| 1.1.1.1.9 US IND Annual Report, Date: | |
| 1.1.1.1.10 | |
| 1.1.1.1.11 | |
| 1.1.1.1.12 | ) |
| Total # of pages in this transmission, including coverpage: | |